# A Phase 2 Study of Check Point Inhibitor, Durvalumab (MEDI4736) for Bacillus Calmette-Guérin (BCG) Refractory Urothelial Carcinoma in Situ (CIS) of the Bladder

NCT02901548

Version 1.9.4

June 12, 2019

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

Investigational Drug

Substance(s)

Durvalumab (Medi4736)

Study Number

MCC18788/ESR-15-11326

Version Number

1.9.4

Date

06/12/2019

A phase 2 study of check point inhibitor, Durvalumab (MEDI4736) for bacillus Calmette-Guérin (BCG) refractory urothelial carcinoma in situ (CIS) of the bladder

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4
Date 06/12/2019

# STUDY PERSONNEL

| Sponsor: | H Lee Moffitt Cancer Center 12902 Magnolia Drive Tampa EL 22(12) |
|---|---|
| | Tampa, FL 33612 |
| Study Location: | H. Lee Moffitt Cancer Center and Research Institute |
| Principal Investigator: | Jingsong Zhang, M.D., Ph.D. |
| Timelpai investigator. | 12902 Magnolia Dr. |
| | Tampa, FL 33612 |
| | Tel: 813 745 1363 |
| | Fax: 813 745 8494 |
| | Email: jingsong.zhang@moffitt.org |
| Co-Investigators | Wade Sexton, M.D., Scott Gilbert M.D., Michael Poch, |
| Co-investigators | M.D., Julio Pow-Sang, M.D., Philippe Spiess M.D. |
| | Biostatistician |
| | Youngchul Kim, Ph.D |

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

# PROTOCOL SYNOPSIS

# Clinical Protocol: MCC18788/ ESR-15-11326

**Study Title:** A phase 2 study of check point inhibitor, Durvalumab (MEDI4736) for Bacillus Calmette-Guérin (BCG) refractory urothelial carcinoma in situ (CIS) of the bladder

Protocol Number: MCC18788/ ESR-15-11326

Clinical Phase: phase 2

**Study Duration: 3-4 years** 

#### **Investigational Product(s) and Reference Therapy:**

Durvalumab will be supplied in glass vials containing 500 mg of liquid solution at a concentration of 50 mg/mL for intravenous (IV) administration.

# **Research Hypothesis:**

Durvalumab will be effective in treating BCG refractory urothelial CIS of bladder

# **Objectives:**

# **Primary Objectives:**

To evaluate whether Durvalumab can improve complete response rate at month 6 to 40% or higher

# **Secondary Objective(s)**:

To evaluate whether Durvalumab can improve the response rate at year 2 to 30% or higher. To assess the safety and tolerability of Durvalumab at 1500 mg Q4W IV infusion for 12 months.

# **Exploratory Objective(s):**

- Correlate PD-L1 expression in urothelial carcinoma, tumor infiltrating T cells, mononuclear cells in bladder biopsies or TURBT samples with response to Durvalumab
- Correlate chromosomal abnormalities detected by UroVysion urine test with response to Durvalumab
- Compare the tumor mutation burden and alterations in DNA repair genes in the pre and post Durvalumab urothelial bladder cancer samples

#### **Study Design:**

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

This is a multicenter, open-label, Phase 2 study of Durvalumab to evaluate its antitumor activity for BCG refractory urothelial carcinoma in situ (CIS) of the bladder. Durvalumab will be given every 4 weeks at 1500 mg IV for total of 12 months. Cystoscopy with biopsy and TURBT (if indicated) will be performed at baseline, and every 3 months during the 12 months treatment period and then every 4 months in the 12 month surveillance period. Of note, cystoscopy at baseline, month 6, and 24 will be performed in the operating room with mapping biopsies. Patients will be off study if any of the biopsies document muscle invasive (T2 or above) urothelial carcinoma. Patients will also be off study if their month 6, 12, 16, 20, biopsies show persistent (month 6) or recurrent CIS or invasive (T1 or above) urothelial carcinoma. Otherwise, patients will remain on study until after the month 24 biopsy.

Number of Centers: 2-3 centers in North America

**Number of Subjects: 34** 

# **Study Population:**

Adult male or female subjects with pathologically confirmed urothelial carcinoma in situ (CIS) of the bladder that is refractory to BCG (see inclusion criteria 2).

#### **Inclusion Criteria:**

- 1. Age  $\geq$  18 years at the time of screening with life expectancy of  $\geq$  2 years
- 2. Must have pathologically confirmed urothelial carcinoma in situ (CIS) of the bladder that meet one of the following criteria:
  - 1. Persistence of high-grade CIS at 6 months following an adequate course of BCG; OR
  - 2. Stage/grade progression at 3 months after induction BCG; OR
  - 3. Recurrence of high-grade CIS after achieving a disease-free state (i.e., CR) following induction of an adequate course of BCG that occurs < 9 months after the last exposure to BCG; OR
  - 4. Persistent CIS noted on the bladder biopsies within 3 months of completing at least 2 induction BCG (minimum of five weekly instillations).

An adequate course of BCG should be defined as at least one course of induction (minimum of five weekly instillations) and one maintenance (two of three instillations) in a 6 months period, with an exception for any patient with grade/stage progression after induction BCG (minimum of five weekly instillations).

3. ECOG performance status of 0-1.

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

- 4. Adequate organ and marrow function, as defined as:
  - Hemoglobin  $\geq 9.0 \text{ g/dL}$ ,
  - Absolute neutrophil count (ANC)  $\geq 1.5 \times 10^9 / L (\geq 1500 \text{ per mm}^3)$ ,
  - Platelet count  $\ge 100 \text{ x } 10^9/\text{L } (\ge 100,000 \text{ per mm}^3)$
  - AST (SGOT)/ALT (SGPT)  $\leq 2.5$  x institutional upper limit of normal
  - Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL = Weight (kg) x 
$$(140 - Age)$$
.  
(mL/min) =  $72 \times \text{measure} \text{$ 

Females:

- 5. Written informed consent and any locally required authorization (e.g., HIPAA in the USA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
- 6. Female subjects must not be pregnant, or breast feeding and must have a negative urine or serum pregnancy test within 28 days prior to treatment on Day 1. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 90 days after the final dose of Durvalumab. They must also refrain from egg cell donation for 90 days after the final dose of Durvalumab.
- 7. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception and refrain from sperm donation from Day 1 through 90 days after receipt of the final dose of Durvalumab.

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

#### **Exclusion Criteria:**

- 1. Muscle invasive (T2 or above) urothelial carcinoma or urothelial carcinoma outside the bladder.
- 2. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) or previous enrolment in the present study.
- 3. Participation in another clinical study with an investigational product during the last 4 weeks.
- 4. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
- 5. History of another primary malignancy except for:
  - Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence.
  - Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  - Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ.
- 6. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, tyrosine kinase inhibitor, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent)  $\leq 30$  days prior to the first dose of study drug and within 6 weeks for nitrosourea, mitomycin C or intravesicle therapy).
- 7. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
- 8. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
- 9. Any unresolved toxicity (CTCAE grade 2 or above) from previous anti-cancer

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

# therapy.

- 10. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
- 11. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
- 12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
- 13. History of primary immunodeficiency.
- 14. History of allogeneic organ transplant.
- 15. History of pneumonitis.
- 16. History of hypersensitivity to durvalumab or any excipient.
- 17. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject with confirmed acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
- 18. Known history of previous clinical diagnosis of tuberculosis.
- 19. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
- 20. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
- Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
- 22. Subjects with uncontrolled seizures.

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

23. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.

# **Investigational Product(s), Dose and Mode of Administration:**

Durvalumab will be given at 1500 mg Q4W (equivalent to 20 mg/kg Q4W) IV infusion for 12 months. Population PK analysis indicated only minor impact of body weight (WT) on PK of durvalumab (coefficient of  $\leq 0.5$ ). Please refer to fixed dose under 1.2.2 for details.

# **Study Assessments and Criteria for Evaluation:**

**Safety Assessments:** Adverse events and toxicity will be captured with CTCAE version 4.03. Based on the generally healthy condition of patients with stage 0 is or stage I (with Cis component), we do not anticipate significant toxicities. The study will also be stopped early if 3 or more subjects in the first 10 subjects developed SAEs attributed to Durvalumab.

# **Efficacy Assessments:**

Complete response rate at month 6 as determined by mapping biopsy at month 6 during treatment with Durvalumab.

Complete response rate at year 2 as determined by mapping biopsy at year 2 after 1 year of Durvalumab.

#### **Statistical Methods and Data Analysis:**

Statistical analysis for the primary and secondary endpoints will be descriptive.

Sample Size Determination: The null hypothesis is the 18% historical complete response rate at month 6 will be tested against a one-sided alternative of 40% or higher complete response rate with Durvalumab at month 6 in BCG refectory CIS of bladder. We use a Simon's two-stage design (Simon, 1989) based on the optimal two-stage designs and admissible designs (Jung et al. 2004) for Phase II single arm clinical trials. The required total number of subjects is 34. 13 is the number of subjects accrued during stage 1. If 3 or fewer responses are observed during stage 1, the trial is stopped early for futility. If 9 or fewer responses of total 34 patients are observed by the end of stage two, then no further investigation of the drug is warranted. This design yields a one-sided type I error rate of 0.047 and power of 80% when the true response rate is 40% based on Simon's optimal two-stage design.

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

# SCHEDULE OF STUDY ASSESSMENTS

# Schedule of study assessments: Screening and Treatment Period (<<12 months: maximum of 13 doses, last infusion week 50>>)

| | | All asses | sments to be performed | pre-infusion unless | stated otherwis | se |
|---|---|---|---|---|---|---|
| Assessments to be performed at the times stipulated in the table and as clinically required in the management of the subject. | Screening | 1 | Every 4 weeks | Every 3 months of 12 months treatment phase | Every 4<br>months of the<br>12 months<br>surveillance<br>phase | End of Trial<br>visit |
| Day | -28 to -1 | 1 | Day 1 of the week | | | |
| Week | -4 to -1 | 0 | 4, 8, 12,16, 20, 24, 28,<br>32, 36, 40, 44, 48, | 14, 26, 38, 52 | 68, 86 104, | 105 |
| | | | (± 3 days) | (± 14 days) | (±14 days) | (±7 days) |
| Written informed<br>consent/assignment<br>of subject<br>identification<br>number | X | | | | | |
| Demography and history of tobacco and alcohol use | X | | | | | |
| Previous treatments for CIS of bladder | X | | | | | |
| Formal verification of eligibility criteria | X | | | | | |
| Hepatitis B and C;<br>HIV | X | | | | | |
| Urine hCG or serum βhCG <sup>b</sup> | X | As clinica | ally indicated | - | | - |
| Durvalumab<br>administration | | X | X | | | |
| Clinic visit with<br>history and physical<br>examination <sup>c</sup> | X | X | X | | X | X |

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

# Schedule of study assessments: Screening and Treatment Period (<<12 months: maximum of 13 doses, last infusion week 50>>)

| | | All asses | sments to be performed | pre-infusion unless | stated otherwis | e |
|---|---|---|---|---|---|---|
| Assessments to be performed at the times stipulated in the table and as clinically required in the management of the subject. | Screening | | Every 4 weeks | Every 3 months of 12 months treatment phase | Every 4<br>months of the<br>12 months<br>surveillance<br>phase | End of Trial<br>visit |
| Day | -28 to -1 | 1 | Day 1 of the week | • | | |
| Week | -4 to -1 | 0 | 4, 8, 12,16, 20, 24, 28,<br>32, 36, 40, 44, 48, | 14, 26, 38, 52 | 68, 86 104, | 105 |
| | | | (± 3 days) | (± 14 days) | (±14 days) | (±7 days) |
| Vital signs (pre-<br>during and post-<br>infusion vital signs<br>assessments) <sup>d</sup> | X | X | X | X | X | X |
| Electrocardiogram <sup>e</sup> | X | X then<br>as<br>clinically<br>indicated | | | | |
| Adverse event/serious adverse event assessment | X | X | All visits | | | |
| Concomitant medications | X | X | All visits | | | |
| ECOG performance status | X | X | X | | X | |
| Liver enzyme panelf | | | X | | X | |
| Serum Chemistry (complete clin chem. panel including Liver enzymes, amylase and lipase) <sup>f</sup> | X | X | X | | | |
| Thyroid function<br>tests (TSH and fT3<br>and fT4) <sup>g</sup> | X | X | X | | X | |
| Hematology <sup>f</sup> | X | X | X | | X | |
| Urinalysis <sup>h</sup> | X | | X | | | |

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

Edition Number 1.9.4 Date 06/12/2019

# Schedule of study assessments: Screening and Treatment Period (<<12 months: maximum of 13 doses, last infusion week 50>>)

| | | All assess | sments to be performed | pre-infusion unless | stated otherwis | e |
|---|---|---|---|---|---|---|
| Assessments to be performed at the times stipulated in the table and as clinically required in the management of the subject. | Screening | 1 | Every 4 weeks | Every 3 months of 12 months treatment phase | Every 4<br>months of the<br>12 months<br>surveillance<br>phase | End of Trial<br>visit |
| Day | -28 to -1 | 1 | Day 1 of the week | 1 | | ı |
| Week | -4 to -1 | 0 | 4, 8, 12,16, 20, 24, 28,<br>32, 36, 40, 44, 48, | 14, 26, 38, 52 | 68, 86 104, | 105 |
| | | (± 3 days) | (± 14 days) | (±14 days) | (±7 days) | |
| Coagulation parameters <sup>i</sup> | X | As clinica | ally indicted | | | |
| Cystoscopy with biopsy <sup>j</sup> | X | | | X | X | |
| Urine cytology with<br>UroVysion test | X | | | X at week 26 | X at week 104 | |
| Tumor assessment<br>(chest X-ray,<br>abdominal pelvic<br>CT) <sup>k</sup> | X | | | | | |

<sup>&</sup>lt;sup>a</sup> Within the protocol could state if for that trial there is a minimum number of subjects to be sampled

- At the beginning of the infusion (at 0 minutes)
- At 30 minutes during the infusion ( $\pm 5$  minutes)
- At the end of the infusion (at 60 minutes  $\pm 5$  minutes)
- In the 1 hour observation period post-infusion: 30 and 60 minutes after the infusion (ie, 90 and 120 minutes from the start of the infusion) (±5 minutes) for the first infusion only and then for subsequent infusions as clinically indicated If the infusion takes longer than 60 minutes then blood pressure and pulse measurements should be collected every 30 minutes (±5 minutes) and as described above or more frequently if clinically indicated.
- e ECG during screening and at Day1 –baseline. There after as clinically indicated. Baseline and abnormal ECG at any time in triplicate others single. 1 ECG is needed while on treatment>>, and as clinically indicated. ECGs should be taken within an hour prior to the start of the infusion and at least one time point 0 to 3 hours after the infusion.
- f If screening laboratory assessments are performed within 3 days prior to Day 1 they do not need to be repeated at Day 1. Results for safety bloods must be available and reviewed before commencing an infusion. Gamma glutamyltransferase tested at Screening, Day 1 and as clinically indicated.

<sup>&</sup>lt;sup>b</sup> Pre-menopausal female subjects of childbearing potential only

<sup>&</sup>lt;sup>e</sup> Full physical examination at baseline; targeted physical examination (including weight and vital signs) at other timepoints

<sup>&</sup>lt;sup>d</sup> Subjects will have their blood pressure and pulse measured before, during and after the infusion at the following times (based on a 60-minute infusion):

Drug Substance Durvalumab (Medi4736) Study Number: MCC 18788/ESR-15-11326

- g Free T3 and free T4 will only be measured if TSH is abnormal. They should also be measured if there is clinical suspicion of an adverse event related to the endocrine system.
- h Urinalysis performed at Screening, Day 1, every 4 weeks and as clinically indicated.
- i Coagulation tests: prothrombin time, APTT and INR only performed at Screening and as clinically indicated.
- j Cystoscopy at baseline, week 26/month 6, and week 104/month 24 will be performed in the operating room with mapping biopsies. The mapping biopsy at baseline can be waived if the subject has a cystoscopy within 8 weeks, which documented recurrent or persistent CIS without evidence of muscle invasive urothelial bladder cancer. After month 3, 9, 12, 16 and 20 cystoscopy, a biopsy will be performed at the discretion of the Urologist.
- k Chest X-ray and CT (preferably with IV contrast) are collected during screening (for baseline) to rule out metastatic disease and secondary malignancy, Due to the low risk of metastasis with CIS of bladder, repeat imaging studies will not be indicated until cancer in the bladder has progressed to the muscle invasive stage. At this point subjects will be off study due to disease progression

| TABLE OF CONTENTS | | |
|---|---|---|
| | SYNOPSIS | 3 |
| | SCHEDULE OF ASSESSMENTS | 9 |
| | TABLE OF CONTENTS | 13 |
| | ABBREVIATIONS AND DEFINITION OF TERMS | 19 |
| 1. | INTRODUCTION | 24 |
| 1.1 | Disease Background | 24 |
| 1.2 | Durvalumab Background | 25 |
| 1.2.1 | Summary of non-clinical experience | 25 |
| 1.2.2 | Summary of clinical experience | 27 |
| 1.3 | Research hypothesis | 31 |
| 1.4 | Rationale for conducting this study | 31 |
| 1.5 | Benefit/risk and ethical assessment | 32 |
| 2. | STUDY OBJECTIVES | 33 |
| 2.1 | Primary objective(s) | 33 |
| 2.2 | Secondary objective(s) | 33 |
| 2.3 | Exploratory objective(s) | 33 |
| 3. | STUDY DESIGN | 33 |
| 3.1 | Overview of study design | 33 |
| 3.2 | Study schema | 34 |
| 3.3 | Study Oversight for Safety Evaluation | 36 |
| 4. | SUBJECT SELECTION | 36 |
| 4.1 | Inclusion criteria | 36 |
| 4.2 | Exclusion criteria | 37 |
| 4.3 | Withdrawal of Subjects from Study Treatment and/or Study | 40 |
| 4.4 | Replacement of subjects | 41 |
| 5. | INVESTIGATIONAL PRODUCT(S) | 41 |

Edition Number 1.9.4

Date 10/08/2018

| 5.1 | Durvalumab | 41 |
|---|---|---|
| 5.1.1 | Formulation/packaging/storage | 41 |
| 5.1.2 | Durvalumab Doses and treatment regimens | 41 |
| 5.1.3 | Study drug preparation | 42 |
| 5.1.4 | Monitoring of dose administration | 43 |
| 5.1.5 | Accountability and dispensation | 44 |
| 5.1.6 | Disposition of unused investigational study drug | 44 |
| 6. | TREATMENT PLAN | 45 |
| 6.1 | Subject enrollment | 45 |
| 6.2 | Dosage and Administration | 45 |
| 6.3 | Dose Modification and Toxicity Management | 45 |
| 7. | RESTRICTIONS DURING THE STUDY AND CONCOMITANT | |
| | TREATMENT(S) | 47 |
| 7.1 | Restrictions during the study | 47 |
| 7.2 | Concomitant treatment(s) | 48 |
| 7.2.1 | Permitted concomitant medications | 48 |
| 7.2.2 | Excluded Concomitant Medications | 48 |
| 8. | STUDY PROCEDURES | 49 |
| 8.1 | Schedule of study procedures | 49 |
| 8.1.1 | Screening Phase | 49 |
| 8.1.2 | Treatment Phase | 50 |
| 8.1.3 | End of Treatment | 50 |
| 8.2 | Description of study procedures | 51 |
| 8.2.1 | Medical history and physical examination, electrocardiogram, weight and | |
| | vital signs | 51 |
| 8.2.2 | Clinical laboratory tests | 52 |
| 8.3 | Biological sampling procedures | 54 |
| 9. | DISEASE EVALUATION AND METHODS | 58 |
| 9.1.1 | Pathological response | 60 |

| 9.1.2 | Urine cytology and UroVysion test6 | |
|---|---|---|
| 10. | ASSESSMENT OF SAFETY | 59 |
| 10.1.1 | Safety Parameters | 59 |
| 10.1.1.1 | Definition of adverse events | 59 |
| 10.1.2 | Definition of serious adverse events | 60 |
| 10.1.3 | Definition of adverse events of special interest (AESI) | 60 |
| 10.1.4 | Pneumonitis | 61 |
| 10.1.5 | Hypersensitivity Reactions | 61 |
| 10.1.6 | Hepatic function abnormalities (hepatotoxicity) | 62 |
| 10.1.7 | Gastrointestinal disorders | 62 |
| 10.1.8 | Endocrine disorders | 63 |
| 10.1.9 | Pancreatic disorders | 63 |
| 10.1.10 | Neurotoxicity | 63 |
| 10.1.11 | Nephritis | 63 |
| 10.2 | Assessment of safety parameters | 64 |
| 10.2.1 | Assessment of severity | 64 |
| 10.2.2 | Assessment of relationship | 65 |
| 10.3 | Recording of adverse events and serious adverse events | 65 |
| 10.3.1 | Study recording period and follow-up for adverse events and serious | |
| | adverse events | 66 |
| 10.3.2 | Reporting of serious adverse events | 67 |
| 10.3.3 | Reporting of deaths | 68 |
| 10.3.4 | Other events requiring reporting | 69 |
| 10.3.5 | Overdose | 69 |
| 10.3.6 | Hepatic function abnormality | 69 |
| 10.3.7 | Pregnancy | 70 |
| 10.3.8 | Maternal exposure | 70 |
| 10.3.9 | Paternal exposure | 71 |
| 11. | STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION | 71 |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

| 11.1 | Description of analysis sets | 71 |
|---|---|---|
| 11.1.1 | Safety analysis set | 71 |
| 11.1.2 | Efficacy analysis set | 71 |
| 11.2 | Methods of statistical analyses | 72 |
| 11.2.1 | Safety Analyses | 72 |
| 11.2.2 | Efficacy Analyses | 73 |
| 11.2.3 | Exploratory Analyses | 73 |
| 11.2.4 | Interim analyses | 73 |
| 11.3 | Determination of sample size | 73 |
| 12. | ETHICAL AND REGULATORY REQUIREMENTS | 73 |
| 12.1 | Ethical conduct of the study | 73 |
| 12.2 | Ethics and regulatory review | 74 |
| 12.3 | Informed consent | 74 |
| 12.4 | Changes to the protocol and informed consent form | 75 |
| 12.5 | Audits and inspections | 75 |
| 13. | STUDY MANAGEMENT | 75 |
| 13.1 | Training of study site personnel. | 75 |
| 13.2 | Monitoring of the study | 75 |
| 13.3 | Study timetable and end of study | 76 |
| 13.4<br>14. | Affiliate Sites Required Documentation. DATA MANAGEMENT | |
| 14.1<br>14.2 | Data Management and Monitoring/Auditing. Study governance and oversight | 77 |
| 15. | INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS | 78 |
| 15.1 | Identity of investigational product(s) | 78 |
| 16 | LIST OF REFERENCES | 78 |

Edition Number 1.9.4
Date 10/08/2018

# LIST OF TABLES

| Table 1 | Dose Modifications and Toxicity Management Guidelines for Immune-Mediated Reactions Associated with Durvalumab82 |
|---|---|
| Table 2 | Dosing Modifications and Toxicity Management Guidelines for Infusion-Related Reactions Associated With Durvalumab102 |
| Table 3 | Dosing Modifications and Toxicity Management Guidelines for Non-immune Mediated Reactions Associated With Durvalumab103 |
| Table 4 | Effective methods of contraception (two methods must be used)47 |
| Table 5 | Prohibited and Rescue Medications49 |
| Table 6 | Hematology Laboratory Tests53 |
| Table 7 | Clinical chemistry (Serum or Plasma) Laboratory Tests53 |
| Table 8 | Urinalysis Tests53 |
| Table 9 | List of investigational products for this study78 |
| Figure 1 | Study flow chart |
| LIST OF AP | PPENDICES |
| or Combination | Dosing Modification and Toxicity Management Guidelines for Immune- ion Related, and Non Immune-mediated Reactions (MEDI4736 Monotherapy therapy with Tremelimumab or Tremelimumab monotherapy) November 2017 |
| Appendix B | Durvalumab Dose Calculations |
| Appendix C | Schedule of study procedures: follow-up for subjects who have completed durvalumab treatment and achieved disease control (until confirmed progression of disease) and subjects who have discontinued durvalumab due to toxicity in the absence of confirmed progression of disease105 |

Clinical Study Protocol
Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)
Study Number MCC 18788/MCC18788/ESR-15-11326
Edition Number 1.9.4
Date 10/08/2018

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

# ABBREVIATIONS AND DEFINITION OF TERMS

The following abbreviations and special terms are used in this study Clinical Study Protocol.

| Abbreviation or special term | Explanation |
|------------------------------|-----------------------------------------------|
| ADA | anti-drug antibody |
| ADCC | antibody-dependent cell-mediated cytotoxicity |
| AE | adverse event |
| AESI | adverse event of special interest |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| APC | antigen-presenting cells |
| AST | aspartate aminotransferase |
| AUC | area under the concentration-time curve |
| CDC | Complement dependent cytotoxicity |
| CI | confidence interval |
| CIS | Carcinoma in situ |
| CL | clearance |
| Cmax | peak concentration |
| Cmax,ss | peak concentration at steady state |
| Cmin | trough concentration |
| Cmin,ss | trough concentration at steady state |
| CNS | central nervous system |
| CR | complete response |
| СТ | computed tomography |
| CTLA-4 | cytotoxic T-lymphocyte-associated antigen-4 |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

| Abbreviation or special term | Explanation |
|------------------------------|-------------------------------------------|
| DC | disease control |
| DCR | disease control rate |
| DLT | dose-limiting toxicity |
| DMC | Data monitoring committee |
| DNA | deoxyribonucleic acid |
| DoR | duration of response |
| ECG | electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EDTA | disodium edetate dihydrate |
| Fc | fragment crystallizable |
| FFPE | formalin fixed paraffin embedded |
| FSH | follicle-stimulating hormone |
| FTIH | first-time-in-human |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| GLP | Good Laboratory Practice |
| HC1 | hydrochloride |
| HIV | human immunodeficiency virus |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IFN | interferon |
| IGF | insulin-like growth factor |
| IgG1 | immunoglobulin G1 |
| IgG2 | immunoglobulin G2 |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

| Abbreviation or special term | Explanation |
|---|---|
| IGSF | immunoglobulin superfamily |
| IHC | immunohistochemistry |
| IL | interleukin |
| irAE | immune-related adverse event |
| IRB | Institutional Review Board |
| IV | intravenous(ly) |
| MAb | monoclonal antibody |
| MDSC | Myeloid derived suppressor cells |
| MedDRA | Medical Dictionary for Regulatory Activities |
| miRNA | micro ribonucleic acid |
| MRI | magnetic resonance imaging |
| mRNA | messenger ribonucleic acid |
| MTD | maximum tolerated dose |
| NCI CTCAE | National Cancer Institute Common Terminology Criteria for Adverse<br>Events |
| NK | natural killer |
| NOAEL | no-observed-adverse-effect level |
| NSCLC | non-small cell lung cancer |
| OR | objective response |
| ORR | objective response rate |
| OS | overall survival |
| PBMC | peripheral blood mononuclear cell |
| PD | progressive disease |
| PD-1 | programmed cell death 1 |
| PD-L1 | programmed cell death ligand 1 |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

| Abbreviation or special term | Explanation |
|---|---|
| PD-L2 | programmed cell death ligand 2 |
| PFS | progression-free survival |
| PK | pharmacokinetic(s) |
| PR | partial response |
| PRO | patient-reported outcome |
| PVC | polyvinyl chloride |
| Q2W | every 2 weeks |
| Q3M | every 3 months |
| Q3W | every 3 weeks |
| Q4W | every 4 weeks |
| Q12W | every 12 weeks |
| QoL | quality of life |
| QTc | the time between the start of the Q wave and the end of the T wave corrected for heart rate |
| QTcF | QT interval on ECG corrected using the Frederica's formula |
| RCC | renal cell carcinoma |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SD | stable disease |
| SID | subject identification |
| sPD-L1 | soluble programmed cell death ligand 1 |
| SOCS3 | suppressor of cytokine signaling 3 |
| SUSAR | suspected unexpected serious adverse reaction |
| t½ | half-life |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

| Abbreviation or special term | Explanation |
|------------------------------|----------------------------------------------|
| TEAE | treatment-emergent adverse event |
| TIL | tumor infiltrating lymphocyte |
| Tmax | time to peak concentration |
| Tmax,ss | time to peak concentration at steady state |
| TNF-α | tumor necrosis factor alpha |
| TSH | thyroid stimulating hormone |
| TURBT | transurethral resection of the bladder tumor |
| ULN | upper limit of normal |
| USA | United States of America |
| WFI | water for injection |
| WHO | World Health Organization |

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

# 1. INTRODUCTION

# 1.1 Disease Background

Bladder cancer is the fifth most common cancer in the United States. Approximately 74,690 new cases (56,390 men and 18,300 women) and 15,580 deaths (11,170 men and 4,410 women) from bladder cancer would occur in the United States in 2014. Nearly 75% of newly diagnosed bladder cancers are non-muscle invasive bladder cancer (NMIBC) or "superficial bladder cancer". CIS is a flat high-grade noninvasive urothelial carcinoma (UC) that has a high propensity for invasion and metastasis. It may occur in isolation or with a synchronous UC. Other than bladder, it could also occur in urothelium lines upper tract, prostatic and penile uretheral. The incidence of CIS of bladder is about 14-19% based on the published data with multiple bladder biopsies.

Intravesical BCG remains the most effective treatment for non-muscle invasive bladder cancer. Its efficacy is attributed to immune response induced by BCG, which tends to wane over time. BCG refractory bladder cancer is commonly defined as recurrence after 2 induction courses of BCG, or recurrence within 6 months of completing induction and maintenance phase of BCG. Unlike TURBT for Ta and T1 UC, CIS cannot be completely resected by biopsy. Standard therapy for BCG refractory CIS is radical cystectomy. For patients who are unsuitable for or refuse radical cystectomy, one approach would be enhancing the protective immunity induced by intravesical BCG by adding agents like interferon-α (Lam et al, 2003). Alternative approaches would be intravesical valrubicin or intravesical gemcitabine. Although intravesical valrubicin is the only FDA approved salvage agent, its complete response rate was only 18% at 3 months and 4% at year 2 in BCG refractory or intolerant CIS (Dinney et al, 2013). There is an unmet need to develop more effective therapy for BCG refractory CIS of bladder. Based on the report of the FDA and AUA joint workshop in 2013, an agent with an initial CR rate of 40-50% at month 6 and a durable response rate of at least 30% would be considered meaningful for BCG refractory CIS (Jarow et al, 2014).

Immune responses directed against tumors are one of the body's natural defences against the growth and proliferation of cancer cells. However, over time and under pressure from immune attack, cancers develop strategies to evade immune-mediated killing allowing them to develop unchecked. One such mechanism involves upregulation of surface proteins that deliver inhibitory signals to cytotoxic T cells. Programmed cell death ligand 1 (PD-L1) is one such protein, and is upregulated in a broad range of cancers with a high frequency, with up to 88% expression in some tumor types. In a number of these cancers, including lung (Mu et al, 2011), renal (Thompson et al, 2005; Thompson et al, 2006; Krambeck et al, 2007), pancreatic (Nomi et al, 2007; Loos et al, 2008; Wang et al, 2010), ovarian cancer (Hamanishi et al, 2007), and hematologic malignancies (Andorsky et al, 2011; Brusa et al, 2013) tumor cell expression of PD-L1 is associated with reduced survival and an unfavorable prognosis.

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

Programmed cell death ligand 1 is part of a complex system of receptors and ligands that are involved in controlling T-cell activation. PD-L1 acts at multiple sites in the body to help regulate normal immune responses and is utilized by tumors to help evade detection and elimination by the host immune system tumor response. In the lymph nodes, PD-L1 on antigen-presenting cells binds to PD-1 or CD80 on activated T cells and delivers an inhibitory signal to the T cell (Keir et al, 2008; Park et al, 2010). This results in reduced T-cell activation and fewer activated T cells in circulation. In the tumor microenvironment, PD-L1 expressed on tumor cells binds to PD-1 and CD80 on activated T cells reaching the tumor. This delivers an inhibitory signal to those T cells, preventing them from killing target cancer cells and protecting the tumor from immune elimination (Zou and Chen, 2008).

Previous immunohistochemistry study reported that 45% of CIS expressed PD-L1, which is the highest among different T stages of urothelial carcinoma of the bladder (Inman et al, 2007). In 11 of 12 patients failing BCG treatment, PD-L1 expression was found to be extremely abundant in the BCG-induced bladder granulomata. More recently targeting PD-L1 with MPDL3280A reported activity in metastatic urothelial bladder cancer tumours. The response rate is particularly high in tumours with PD-L1-positive tumour-infiltrating immune cells (Powles et al, 2014). These data support targeting PD-L1 in BCG refractory CIS urothelial bladder cancer.

# 1.2 Durvalumab Background

Durvalumab is being developed as a potential anticancer therapy for patients with advanced solid tumors. Durvalumab is a human monoclonal antibody (MAb) of the immunoglobulin G1 kappa (IgG1κ) subclass that inhibits binding of programmed cell death ligand 1 (PD-L1) (B7 homolog 1 [B7-H1], cluster of differentiation [CD]274) to programmed cell death 1 (PD-1; CD279) and CD80 (B7-1). Durvalumab is composed of 2 identical heavy chains and 2 identical light chains, with an overall molecular weight of approximately 149 kDa. Durvalumab contains a triple mutation in the constant domain of the immunoglobulin (Ig) G1 heavy chain that reduces binding to complement protein C1q and the fragment crystallizable gamma (Fcγ) receptors involved in triggering effector function.

# 1.2.1 Summary of non-clinical experience

Non-clinical experience with durvalumab is fully described in the current version of the durvalumab Investigator's Brochure (Version 12.0)

Durvalumab binds with high affinity and specificity to human PD-L1 and blocks its interaction with PD-1 and CD80. *In vitro* studies demonstrate that durvalumab antagonizes the

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

inhibitory effect of PD-L1 on primary human T cells, resulting in their restored proliferation and release of interferon gamma (IFN- $\gamma$ ). Additionally, durvalumab demonstrated a lack of antibody-dependent cell-mediated cytotoxicity (ADCC) and complement-dependent cytotoxicity (CDC) in cell-based functional assays. In vivo studies show that durvalumab inhibits tumor growth in a xenograft model via a T lymphocyte (T-cell) dependent mechanism. Moreover, an anti-mouse PD-L1 antibody demonstrated improved survival in a syngeneic tumor model when given as monotherapy and resulted in complete tumor regression in > 50% of treated mice when given in combination with chemotherapy. Combination therapy (dual targeting of PD-L1 and cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4]) resulted in tumor regression in a mouse model of colorectal cancer.

Cynomolgus monkeys were selected as the only relevant species for evaluation of the pharmacokinetics (PK)/pharmacodynamics and potential toxicity of durvalumab. Following intravenous (IV) administration, the PK of durvalumab in cynomolgus monkeys was nonlinear. Systemic clearance (CL) decreased and concentration half-life (t1/2) increased with increasing doses, suggesting saturable target binding-mediated clearance of durvalumab. No apparent gender differences in PK profiles were observed for durvalumab.

In general, treatment of cynomolgus monkeys with durvalumab was not associated with any durvalumab -related adverse effects that were considered to be of relevance to humans. Adverse findings in the non-Good Laboratory Practice (GLP) PK/pharmacodynamics and dose range-finding study, and a GLP 4-week repeat-dose toxicity study were consistent with antidrug antibody (ADA)-associated morbidity and mortality in individual animals. The death of a single animal in the non-GLP, PK/pharmacodynamics, and dose range-finding study was consistent with an ADA-associated acute anaphylactic reaction. The spectrum of findings, especially the clinical signs and microscopic pathology, in a single animal in the GLP, 4-week, repeat-dose study was also consistent with ADA immune complex deposition, and ADA: durvalumab immune complexes were identified in a subsequent non-GLP, investigative immunohistochemistry study. Similar observations were reported in cynomolgus monkeys administered human mAbs unrelated to durvalumab. Given that immunogenicity of human mAbs in nonclinical species is generally not predictive of responses in humans, the ADA-associated morbidity and mortality were not considered for the determination of the no-observed-adverse-effect level (NOAEL) of durvalumab.

Finally, data from the pivotal 3-month GLP toxicity study with durvalumab in cynomolgus monkeys showed that subchronic dosing of durvalumab was not associated with any adverse effects. Therefore, the NOAEL of durvalumab in all the general toxicity studies was considered to be 100 mg/kg, the highest dose tested in these studies. In addition to the *in vivo* 

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

toxicology data, no unexpected membrane binding of durvalumab to human or cynomolgus monkey tissues was observed in GLP tissue cross-reactivity studies using normal human and cynomolgus monkey tissues.

# 1.2.2 Summary of clinical experience

Clinical experience with durvalumab is fully described in the current version of the durvalumab Investigator's Brochure (Version 12.0).

As of the DCO dates (15Apr2015 to 12Jul2015, Durvalumab IB Version 9.0), a total of 1,883 subjects have been enrolled and treated in 30 ongoing durvalumab clinical studies, including 20 sponsored and 10 collaborative studies. Of the 1,883 subjects, 1,279 received durvalumab monotherapy, 440 received durvalumab in combination with tremelimumab or other anticancer agents, 14 received other agents (1 gefitinib, 13 MEDI6383), and 150 have been treated with blinded investigational product. No studies have been completed or terminated prematurely due to toxicity.

#### Pharmacokinetics and Product Metabolism

Study CD-ON-durvalumab-1108: As of 09 Feb2015, PK data were available for 378 subjects in the dose-escalation and dose-expansion phases of Study CD-ON-durvalumab-1108 following treatment with durvalumab 0.1 to 10 mg/kg every 2 weeks (Q2W) or 15 mg/kg every 3 weeks (Q3W). The maximum observed concentration ( $C_{max}$ ) increased in an approximately dose-proportional manner over the dose range of 0.1 to 15 mg/kg. The area under the concentration-time curve from 0 to 14 days (AUC<sub>0-14</sub>) increased in a greater than dose-proportional manner over the dose range of 0.1 to 3 mg/kg and increased dose-proportionally at  $\geq$  3 mg/kg. These results suggest durvalumab exhibits nonlinear PK likely due to saturable target-mediated CL at doses < 3 mg/kg and approaches linearity at doses  $\geq$  3 mg/kg. Near complete target saturation (soluble programmed cell death ligand 1 [sPD-L1] and membrane bound) is expected with durvalumab  $\geq$  3 mg/kg Q2W. Exposures after multiple doses showed accumulation consistent with PK parameters estimated from the first dose. In addition, PK simulations indicate that following durvalumab 10 mg/kg Q2W dosing, > 90% of subjects are expected to maintain PK exposure  $\geq$  40  $\mu$ g/mL throughout the dosing interval.

As of 09 Feb2015, a total of 388 subjects provided samples for ADA analysis. Only 8 of 388 subjects (1 subject each in 0.1, 1, 3, and 15 mg/kg cohorts, and 4 subjects in 10 mg/kg cohort) were ADA positive with an impact on PK/pharmacodynamics in 1 subject in the 3 mg/kg cohort.

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

#### Safety

The safety profile of durvalumab as monotherapy and combined with other anticancer agents was consistent with the pharmacology of the target and other agents in the immune checkpoint inhibitor class. No tumor types appeared to be associated with unique AEs. Immune-related AEs (irAEs), which are important risks of immune checkpoint inhibitors, have been observed with durvalumab and include colitis, pneumonitis, hepatitis/hepatotoxicity, neuropathy/neuromuscular toxicity, endocrinopathy, dermatitis, and nephritis. In addition, pancreatitis is an important potential risk particularly with durvalumab and tremelimumab combination therapy. These events are manageable by available/established treatment guidelines as described in the study protocols.

AEs reported with durvalumab monotherapy in key clinical studies are described below.

# **Adverse Event Profile of durvalumab Monotherapy**

Study CD-ON-durvalumab-1108: The safety profile of durvalumab monotherapy in the 694 subjects with advanced solid tumors treated at 10 mg/kg Q2W in Study CD-ON-durvalumab-1108 has been broadly consistent with that of the overall 1,279 subjects who have received durvalumab monotherapy (not including subjects treated with blinded investigational product) across the clinical development program. The majority of treatmentrelated AEs were manageable with dose delays, symptomatic treatment, and in the case of events suspected to have an immune basis, the use of established treatment guidelines for immune-mediated toxicity. As of 07 May2015, among the 694 subjects treated with durvalumab 10 mg/kg Q2W in Study CD-ON-durvalumab-1108, a total of 378 subjects (54.5%) experienced a treatment-related AE, with the most frequent (occurring in  $\geq$  5% of subjects) being fatigue (17.7%), nausea (8.6%), diarrhea (7.3%), decreased appetite (6.8%), pruritus (6.3%), rash (6.1%), and vomiting (5.0%). A majority of the treatment-related AEs were Grade 1 or Grade 2 in severity with  $\geq$  Grade 3 events occurring in 65 subjects (9.4%). Treatment-related  $\geq$  Grade 3 events reported in 3 or more subjects ( $\geq$  0.4%) were fatigue (12 subjects, 1.7%); increased aspartate aminotransferase (AST; 7 subjects, 1.0%); increased gamma-glutamyltransferase (GGT; 6 subjects, 0.9%); increased alanine aminotransferase (ALT; 5 subjects, 0.7%); and colitis, vomiting, decreased appetite, and hyponatremia (3 subjects, 0.4% each). Six subjects had treatment-related Grade 4 AEs (upper gastrointestinal hemorrhage, increased AST, dyspnea, neutropenia, colitis, diarrhea, and pneumonitis) and 1 subject had a treatment-related Grade 5 event (pneumonia). Treatmentrelated serious adverse events (SAEs) that occurred in  $\geq 2$  subjects were colitis and pneumonitis (3 subjects each). A majority of the treatment-related SAEs were ≥ Grade 3 in

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

severity and resolved with or without sequelae. AEs that resulted in permanent discontinuation of durvalumab were considered as treatment related in 18 subjects (2.6%), with colitis being the most frequent treatment-related AE resulting in discontinuation (3 subjects). A majority of the treatment-related AEs resulting in discontinuation of durvalumab were  $\geq$  Grade 3 in severity and resolved with or without sequelae.

Study D4191C00003/ATLANTIC: The safety profile of durvalumab monotherapy in consistent Study CD-ON-durvalumab-1108 is generally with that of Study D4191C00003/ATLANTIC in subjects with locally advanced or metastatic non-smallcell lung cancer (NSCLC) treated with durvalumab 10 mg/kg O2W. As of 05May2015, 264 of 303 subjects (87.1%) reported any AE in Study D4191C00003/ATLANTIC. Overall, events reported in  $\geq 10\%$  of subjects were dyspnea (18.8%), fatigue (17.8%), decreased appetite (17.5%), cough (14.2%), pyrexia (12.2%), asthenia (11.9%), and nausea (11.2%). Nearly twothirds of the subjects experienced AEs that were Grade 1 or 2 in severity and manageable by general treatment guidelines as described in the current durvalumab study protocols. Grade 3 or higher AEs were reported in 107 of 303 subjects (35.3%). A total of 128 subjects (42.2%) reported AEs that were considered by the investigator as related to investigational product. Treatment-related AEs (all grades) reported in ≥ 2% of subjects were decreased appetite (6.6%); fatigue (5.9%); asthenia (5.0%); nausea (4.6%); pruritus (4.3%); diarrhea, hyperthyroidism, hypothyroidism, and pyrexia (3.3% each); rash (2.6%); weight decreased (2.3%); and vomiting (2.0%). Treatment-related Grade 3 AEs reported in  $\geq 2$  subjects were pneumonitis (3 subjects) and increased GGT (2 subjects). There was no treatment-related Grade 4 or 5 AEs. Ninety-four of 303 subjects (31.0%) reported any SAE. SAEs that occurred in  $\geq 1.0\%$  of subjects were dyspnea (6.6%); pleural effusion, general physical health deterioration (2.3% each); pneumonia (2.0%); hemoptysis, pulmonary embolism (1.3% each); and pneumonitis, respiratory failure, disease progression (1.0% each). Nine subjects had an SAE considered by the investigator as related to durvalumab. Each treatment-related SAE occurred in 1 subject each with the exception of pneumonitis, which occurred in 3 subjects. Fifteen of 303 subjects (5.0%) have died due to an AE (pneumonia [3 subjects]; general physical health deterioration, disease progression, hemoptysis, dyspnea [2 subjects each]; pulmonary sepsis, respiratory distress, cardiopulmonary arrest [verbatim term (VT)], hepatic failure, and sepsis [1 subject each]). None of these events was considered related to durvalumab. Twenty-three of 303 subjects (7.6%) permanently discontinued durvalumab treatment due to AEs. Events that led to discontinuation of durvalumab in  $\geq 2$  subjects were dyspnea, general physical health deterioration, and pneumonia. Treatment-related AEs that led to discontinuation were increased ALT and increased hepatic enzyme, which occurred in 1 subject each.

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

#### **Efficacy**

Study CD-ON-durvalumab-1108: Overall, 456 of 694 subjects treated with durvalumab 10 mg/kg Q2W were evaluable for response (defined as having  $\geq 24$  weeks follow-up, measurable disease at baseline, and  $\geq 1$  follow-up scan, or discontinued due to disease progression or death without any follow-up scan). In PD-L1 unselected patients, the objective response rate (ORR), based on investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, ranged from 0% in uveal melanoma (n = 23) to 20.0% in bladder cancer (n = 15), and disease control rate at 24 weeks (DCR-24w) ranged from 4.2% in triple-negative breast cancer (TNBC; n = 24) to 39.1% in advanced cutaneous melanoma (n = 23). PD-L1 status was known for 383 of the 456 response evaluable subjects. Across the PD-L1-positive tumors, ORR was highest for bladder cancer, advanced cutaneous melanoma, hepatocellular carcinoma (HCC; n = 3 each, 33.3% each), NSCLC (n = 86, 26.7%), and squamous cell carcinoma of the head and neck (SCCHN; n = 22, 18.2%). In the PD-L1-positive subset, DCR-24w was highest in advanced cutaneous melanoma (n = 3, 66.7%), NSCLC (n = 86, 36.0%), HCC and bladder cancer (n = 3 each, 33.3% each), and SCCHN (n = 22, 18.2%).

**Study D4190C00007:** Of the 32 subjects with myelodysplastic syndrome (MDS) treated in Study D4190C00007, 21 subjects had at least 1 post-baseline disease assessment. Among these subjects, the best overall responses were marrow complete remission (mCR) in 4 subjects (19.0%); stable disease (SD) in 4 subjects (19.0%); and progressive disease (PD) in 5 subjects (23.8%). The remaining 8 subjects (38.1%) did not meet the criteria for complete remission (CR), mCR, partial remission (PR), SD, or PD at the date of assessment.

**Study CD-ON-durvalumab-1161:** Of the 65 subjects with metastatic or unresectable melanoma treated with the combination of durvalumab and BRAF inhibitor (BRAFi; dabrafenib)/MEK inhibitor (MEKi; trametinib), 63 subjects were evaluable for response. A total of 35 subjects (55.6%) had a best overall response of confirmed or unconfirmed PR. The disease control rate (DCR; CR + PR [regardless of confirmation] + SD  $\geq$  12 weeks) was 79.4%.

# **Fixed Dosing**

A population PK model was developed for durvalumab using monotherapy data from a Phase 1 study (study 1108; N=292; doses= 0.1 to 10 mg/kg Q2W or 15 mg/kg Q3W; solid tumors). Population PK analysis indicated only minor impact of body weight (WT) on PK of durvalumab (coefficient of  $\leq$  0.5). The impact of body WT-based (10 mg/kg Q2W) and fixed dosing (750 mg Q2W) of durvalumab was evaluated by comparing predicted steady state PK

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

concentrations (5<sup>th</sup>, median and 95<sup>th</sup> percentiles) using the population PK model. A fixed dose of 750 mg was selected to approximate 10 mg/kg (based on median body WT of ~75 kg). A total of 1000 patients were simulated using body WT distribution of 40–120 kg. Simulation results demonstrate that body WT-based and fixed dosing regimens yield similar median steady state PK concentrations with slightly less overall between-subject variability with fixed dosing regimen.

Similar findings have been reported by others [Ng et al 2006, Wang et al. 2009, Zhang et al, 2012, Narwal et al 2013]. Wang and colleagues investigated 12 monoclonal antibodies and found that fixed and body size-based dosing perform similarly, with fixed dosing being better for 7 of 12 antibodies [3]. In addition, they investigated 18 therapeutic proteins and peptides and showed that fixed dosing performed better for 12 of 18 in terms of reducing the between-subject variability in pharmacokinetic/pharmacodynamics parameters [Zhang et al 2012].

A fixed dosing approach is preferred by the prescribing community due to ease of use and reduced dosing errors. Given expectation of similar pharmacokinetic exposure and variability, we considered it feasible to switch to fixed dosing regimens. Based on average body WT of 75 kg, a fixed dose of 750 mg Q2W durvalumab (equivalent to 10 mg/kg Q2W), 1500 mg Q4W durvalumab (equivalent to 20 mg/kg Q4W) is included in the current study. Fixed dosing of durvalumab is recommended only for subjects with > 30kg body weight due to endotoxin exposure. Patients with a body weight less than or equal to 30 kg should be dosed using a weight-based dosing schedule (Appendix B).

# 1.3 Research hypothesis

The null hypothesis that the 18% historical complete response rate at month 6 will be improved to 40% or higher with Durvalumab at month 6 in BCG refectory CIS of bladder. Such hypothesis is supported by the high percentage of PD-L1 IHC positivity in CIS of urothelial bladder cancer and enrichment of PD-L1 expression in the BCG-induced bladder granulomata after BCG failure (Inman et al, 2007). Vascular inflammation induced by bladder mapping biopsy would facilitate the deposition of immune complex containing durvalumab (Investigator brochure) at the biopsy sites.

# 1.4 Rationale for conducting this study

There is an unmet need to develop more effective therapy for BCG refractory CIS of bladder. To facilitate drug development in this disease setting, FDA and AUA held a joint workshop in 2013. Based on the report from this workshop, an agent with an initial CR rate of 40-50% at month 6 and a durable response rate of at least 30% would be considered meaningful for BCG

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

refractory CIS. Response rate at month 6 is chosen as the primary endpoint. The historical 18% month 6 complete response rate will be tested against a one-sided alternative of druvalumab treated patients would show a complete response rate 40% or higher. Response rate at year 2 as well as safety assessments was chosen as secondary objectives.

Durvalumab will be given at 1500 mg Q4W (equivalent to 20 mg/kg Q4W) IV infusion for 12 months. Population PK analysis indicated only minor impact of body weight (WT) on PK of durvalumab (coefficient of  $\leq$  0.5). A fixed dosing approach is preferred due to ease of use and reduced dosing errors.

#### 1.5 Benefit/risk and ethical assessment

As described in section 1.2.2, Durvalumab is well tolerated in human subjects. No tumor types appeared to be associated with unique AEs. Immune-related AEs (irAEs), which are important risks of immune checkpoint inhibitors, have been observed with Durvalumab and include colitis, pneumonitis, hepatitis/hepatotoxicity, neuropathy/neuromuscular toxicity, endocrinopathy, dermatitis, and nephritis. These irAEs are not that different than the anti-PD1or anti-PDL1 agents being approved by FDA for treating melanoma, kidney cancer and non-small cell lung cancer.

Due to the lack of effective intravesical treatment for BCG refractory urothelial carcinoma in situ (CIS) of the bladder, radical cystectomy is often recommended. If subject's CIS of bladder does not respond to IV Durvalumab, delaying cystectomy could lead to cancer progression to the muscle invasive or even metastatic stage. The protocol therefore mandates a baseline staging work up prior to study enrollment and every 3 months cystoscopy with mapping biopsy during the 2 year study period. For subjects who elect bladder preservation for their CIS of bladder, it is a common practice to do every 3 months surveillance cystoscopy till at least a year after completing the intravesical therapy. We don't anticipate adding IV Durvalumab will increase the risks or complications of routine cystoscopy with mapping biopsy. For subjects whose CIS of bladder responded Durvalumab, Durvalumab may provide an alternative treatment that leads to bladder preservation.

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

#### 2. STUDY OBJECTIVES

# 2.1 Primary objective(s)

The primary objective of this study is to evaluate whether Durvalumab can improve complete response rate at month 6 to 40% or above based on the week 26 mapping biopsy in BCG refractory CIS urothelial bladder cancer

# 2.2 Secondary objective(s)

- 1. To evaluate whether Durvalumab can improve the complete response rate at year 2 to 30% or above based on the week 104 mapping biopsy in BCG refractory CIS urothelial bladder cancer
- 2. To assess the safety and tolerability of Durvalumab at 1500 mg Q4W IV infusion for 12 months for BCG refractory CIS urothelial bladder cancer

# 2.3 Exploratory objective(s)

- 1. Correlate PD-L1 expressions in urothelial carcinoma, tumor infiltrating T cells mononuclear cells in bladder biopsy or TURBT samples with response to Durvalumab
- **2.** Correlate chromosomal abnormalities detected by UroVysion urine test with response to Durvalumab
- **3.** Compare the tumor mutation burden and alterations in DNA repair genes in the pre and post Durvalumab urothelial bladder cancer samples

# 3. STUDY DESIGN

# 3.1 Overview of study design

This is a multicenter, open-label, Phase 2 study of Durvalumab to evaluate its antitumor activity for BCG refractory urothelial carcinoma in situ (CIS) of the bladder. We use a Simon's two-stage design (Simon, 1989) based on the optimal two-stage designs and admissible designs (Jung et al. 2004) for Phase II single arm clinical trials. In the first stage of this study plan, 13 patients will be accrued. If there are 3 or fewer responses in these 13 patients, the study will be stopped. Otherwise, 21 additional patients will be accrued for a total of 34. Durvalumab will be given every 4 weeks at 1500 mg IV for total of 12 months/13 doses. Cystoscopy with mapping biopsy and TURBT (if indicated) will be performed at

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

baseline, month 6, and 24. Urine cytology with UroVysion test will be performed at baseline, month 6, and 24. Patients will be off study if any of the biopsies documented muscle invasive (T2 or above) urothelial carcinoma. Patients will also be off study if their month 6, 12, 18 biopsies showed persistent (month 6) or recurrent CIS or invasive (T1 or above) urothelial carcinoma. Otherwise, patient will remain on study until after the month 24 biopsy.

Historical controls will be used to assess the efficacy of Durvalumab. For exploratory analysis on PD-L1 expression, PD-L1 IHC will be performed with the SP263 antibody developed by Ventana. IHC positivity (either on tumor cells and/or infiltrating immune cells) will be assessed on the available mapping biopsy and or TURBT samples at time points defined in SCHEDULE OF STUDY ASSESSMENT.

Data Monitoring Committee (DMC) at Moffitt Cancer Center will monitor this phase 2 study initiated by Moffitt's investigator.

# 3.2 Study schema

Investigational Drug Substance: MEDI4736 Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Figure 1. Study flow chart


Date 10/08/2018

## 3.3 Study Oversight for Safety Evaluation

DMC at Moffitt Cancer Center will monitor this phase 2 study initiated by Moffitt's investigator. The study will be stopped early if there are 3 or fewer responses in the first 13 patients in the stage I of Simon 2 stage design. The study will also be stopped early if 3 or more subjects of the first 10 subjects developed SAEs attributed to Durvalumab.

#### 4. SUBJECT SELECTION

#### 4.1 Inclusion criteria

For inclusion in the study subjects must fulfill all of the following criteria:

- 1. Age  $\geq$  18 years at the time of screening.
- 2. Must have pathologically confirmed urothelial carcinoma in situ (CIS) of the bladder and meet one of the following criteria.
  - 1. Persistence of high-grade CIS at 6 months following an adequate course of BCG; OR
  - 2. Stage/grade progression at 3 months after induction BCG; OR
  - 3. Recurrence of high-grade CIS after achieving a disease-free state (i.e., CR) following induction of an adequate course of BCG that occurs < 9 months after the last exposure to BCG; OR
  - 4. Persistent CIS noted on the bladder biopsies within 3 months of completing at least 2 induction BCG (minimum of five weekly instillations).

An adequate course of BCG should be defined as at least one course of induction (minimum of five weekly instillations) and one maintenance (two of three instillations) in a 6 months period, with an exception for any patient with grade/stage progression after induction BCG (minimum of five weekly instillations).

- 3. ECOG performance status of 0-1.
- 4. Adequate organ and marrow function, as defined as:
  - Haemoglobin  $\geq 9.0$  g/dL, Absolute neutrophil count (ANC)  $\geq 1.5$  x  $10^9$ /L ( $\geq 1500$  per mm<sup>3</sup>), and Platelet count  $\geq 100$  x  $10^9$ /L (>100,000 per mm<sup>3</sup>)

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- AST (SGOT)/ALT (SGPT)  $\leq 2.5$  x institutional upper limit of normal Serum bilirubin  $\leq 1.5$  x institutional upper limit of normal (ULN).
- Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

Creatinine CL = Weight (kg) x (140 - Age) . (mL/min) 72 x serum creatinine (mg/dL)

Females:

Creatinine CL = Weight (kg) x (140 - Age) x 0.85 (mL/min) 72 x serum creatinine (mg/dL)

- 5. Written informed consent and any locally required authorization (e.g., HIPAA in the USA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
- 6. Female subjects must not be pregnant, or breast feeding and must have a negative urine or serum pregnancy test within 28 days prior to treatment on day 1. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 90 days after the final dose of Durvalumab. They must also refrain from egg cell donation for 90 days after the final dose of Durvalumab.
- 7. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception and refrain from sperm donation from Day 1 through 90 days after receipt of the final dose of Durvalumab.

#### 4.2 Exclusion criteria

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- 1. Muscle invasive (T2 or above) urothelial carcinoma or urothelial carcinoma outside the bladder.
- 2. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) or previous enrolment in the present study.
- 3. Participation in another clinical study with an investigational product during the last 4 weeks.
- 4. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab.
- 5. History of another primary malignancy except for:
  - Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence.
  - Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  - Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ.
- 6. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, tyrosine kinase inhibitor, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 30 days prior to the first dose of study drug and within 6 weeks for nitrosourea, mitomycin C or intravesicle therapy).
- 7. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
- 8. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
- 9. Any unresolved toxicity (CTCAE grade 2 or above) from previous anti-cancer therapy. <<Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy)>>

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- 10. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
- 11. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
- 12. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
- 13. History of primary immunodeficiency.
- 14. History of allogeneic organ transplant.
- 15. History of pneumonitis.
- 16. History of hypersensitivity to durvalumab or any excipient.
- 17. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject with confirmed acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
- 18. Known history of previous clinical diagnosis of tuberculosis.
- 19. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
- 20. Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
- 21. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
- 22. Subjects with uncontrolled seizures.
- 23. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.

Edition Number 1.9.4

Date 10/08/2018

## 4.3 Withdrawal of Subjects from Study Treatment and/or Study

#### Permanent discontinuation of Durvalumab

An individual subject will not receive any further investigational product if any of the following occur in the subject in question:

- 1. Withdrawal of consent or lost to follow-up
  - 2. Adverse event that, in the opinion of the investigator or the sponsor, contraindicates further dosing. Patients with grade 3 toxicity at least possibly related to study drug will discontinue durvalumab. Patients with prolonged grade 2 toxicity or who require dose delays for more than 2 weeks or require prolonged steroid use will discontinue durvalumab.
- 3. Subject is determined to have met one or more of the exclusion criteria for study participation at study entry and continuing investigational therapy might constitute a safety risk
- 4. Pregnancy or intent to become pregnant
- 5. Any AE that meets criteria for discontinuation as defined in Appendix A
- 6. Grade > 3 infusion reaction
- 7. Subject noncompliance that, in the opinion of the investigator or sponsor, warrants withdrawal; eg, refusal to adhere to scheduled visits
- 8. Initiation of alternative anticancer therapy including another investigational agent
- 9. Confirmation of PD and investigator determination that the subject is no longer benefiting from treatment with durvalumab

Subjects who are permanently discontinued from further receipt of investigational product, regardless of the reason (withdrawal of consent, due to an AE, other), will be identified as having permanently discontinued treatment.

Subjects who are permanently discontinued from receiving investigational product will be followed for safety per Section 10.3.1 and Appendix C or D, including the collection of any protocol-specified blood specimens, unless consent is withdrawn or the subject is lost to

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

follow-up or enrolled I another clinical study. All subjects will be followed for survival. Subjects who decline to return to the site for evaluations will be offered follow-up by phone every 3 months as an alternative.

#### Withdrawal of consent

If consent is withdrawn, the subject will not receive any further investigational product or further study observation.

## 4.4 Replacement of subjects

Subjects withdrawn from the study prior to the month 6 /week 26 mapping biopsy will be replaced to ensure total of 34 evaluable subjects. Subjects who are incorrectly enrolled but are not yet initiated on treatment should be withdrawn from the study and replaced.

## 5. INVESTIGATIONAL PRODUCT(S)

#### 5.1 Durvalumab

The Investigational Products Supply section of AstraZeneca/MedImmune will supply durvalumab to the investigator as a 500-mg vial solution for infusion after dilution.

#### 5.1.1 Formulation/packaging/storage

Durvalumab will be supplied by AstraZeneca as a 500-mg vial solution for infusion after dilution. The solution contains 50 mg/mL durvalumab, 26 mM histidine/histidine-hydrochloride, 275 mM trehalose dihydrate, and 0.02% (weight/volume) polysorbate 80; it has a pH of 6.0. The nominal fill volume is 10 mL. Investigational product vials are stored at 2°C to 8°C (36°F to 46°F) and must not be frozen. Durvalumab must be used within the individually assigned expiry date on the label.

#### 5.1.2 Durvalumab Doses and treatment regimens

Treatment with fixed dose durvalumab at 1500 mg Q4W durvalumab (equivalent to 20 mg/kg Q4W, based on an average body WT of 75 kg) commences on Day 1 following confirmation of eligibility into the study and continues on a Q4W schedule for a maximum duration of treatment of 12 months (maximum of 13 doses). Study treatment should be discontinued prior to 12 months if there is confirmed PD (unless the investigator considers the subject to continue to receive benefit from treatment), initiation of alternative cancer therapy,

unacceptable toxicity, withdrawal of consent, or if other reasons to discontinue study treatment occur.

Subjects who have a dose interruption due to toxicity at any point in the first 12 months of treatment may resume treatment and complete the 12-month treatment period.

## 5.1.3 Study drug preparation

For patients weighing ≥ 30 kg, 1500 mg Q4W durvalumab (equivalent to 20 mg/kg Q4W) (based on an average body WT of 75 kg) should be prepared. For subjects <30 kg body weight, 20 mg/kg dose should be prepared; dose is determined using body mass, calculating the stock volume of durvalumab to achieve the accurate dose according to Appendix B.

#### Preparation of durvalumab doses for administration with an IV bag

The dose of durvalumab for administration must be prepared by the Investigator's or site's designated IP manager using aseptic technique. Total time from needle puncture of the durvalumab vial to the start of administration should not exceed:

- 24 hours at 2°C to 8°C (36°F to 46°F)
- 4 hours at room temperature

If in-use storage time exceeds these limits, a new dose must be prepared from new vials. Infusion solutions must be allowed to equilibrate to room temperature prior to commencement of administration.

No incompatibilities between durvalumab and polyvinylchloride or polyolefin IV bags have been observed. Dose of 1500mg durvalumab for patients >30 kg will be administered using an IV bag containing 0.9% (w/v) saline with a final durvalumab concentration ranging from 1 to 20 mg/mL, and delivered through an IV administration set with a 0.2- or 0.22- $\mu$ m in-line filter.

Remove a volume of IV solution from the IV bag equal to the calculated volume of durvalumab to be added to the IV bag prior to addition of durvalumab. Next, the volume of durvalumab (ie, 15.0 mL for 750 mg or 30.0 mL for 1500 mg of durvalumab) is added to the IV bag such that final concentration is within 1 to 20 mg/mL (IV bag volumes 100 to 1000 mL). Mix the bag by gently inverting to ensure homogeneity of the dose in the bag.

Patient weight at baseline should be used for dosing calculations in patients  $\leq 30$  kg unless there is a  $\geq 10\%$  change in weight. Dosing day weight can be used for dosing calculations instead of baseline weight per institutional standard.

For patients <30kg, calculate the dose volume of durvalumab and number of vials needed for the subject to achieve the accurate dose according to Appendix B.

Durvalumab will be administered at room temperature (approximately 25°C) by controlled infusion via an infusion pump into a peripheral or central vein. Following preparation of durvalumab, the entire contents of the IV bag should be administered as an IV infusion over approximately 60 minutes (±5 minutes), using a 0.2, or 0.22-μm in-line filter. Less than 55 minutes is considered a deviation.

The IV line will be flushed with a volume of IV solution (0.9% [w/v] saline) equal to the priming volume of the infusion set used after the contents of the IV bag are fully administered, or complete the infusion according to institutional policy to ensure the full dose is administered and document if the line was not flushed.

Standard infusion time is 1 hour. However, if there are interruptions during infusion, the total allowed time should not exceed 8 hours at room temperature. The table below summarizes time allowances and temperatures.

#### **Durvalumab hold and infusion times**

| Maximum time from needle puncture to start of administration | 4 hours at room temperature, 24 hours at 2°C to 8°C |
|---|---|
| Maximum time for IV bag infusion, including interruptions | 8 hours at room temperature |

In the event that either preparation time or infusion time exceeds the time limits outlined above, a new dose must be prepared from new vials. Durvalumab does not contain preservatives, and any unused portion must be discarded.

#### **5.1.4** Monitoring of dose administration

Subjects will be monitored before, during and after the infusion with assessment of vital signs at the times specified in the Schedule of Assessment. Subjects are monitored (pulse rate, blood

pressure) every 30 minutes during the infusion period (including times where infusion rate is slowed or temporarily stopped).

In the event of a ≥Grade 2 infusion-related reaction, the infusion rate of study drug may be decreased by 50% or interrupted until resolution of the event (up to 4 hours) and re-initiated at 50% of the initial rate until completion of the infusion. For subjects with a ≤Grade 2 infusion-related reaction, subsequent infusions may be administered at 50% of the initial rate. Acetaminophen and/or an antihistamine (e.g., diphenhydramine) or equivalent medications per institutional standard may be administered at the discretion of the investigator. If the infusion-related reaction is Grade 3 or higher in severity, study drug will be discontinued. The standard infusion time is one hour, however if there are interruptions during infusion, the total allowed time from infusion start to completion of infusion should not exceed 4 hours at room temperature, with maximum total time at room temperature not exceeding 4 hours (otherwise requires new infusion preparation).

As with any antibody, allergic reactions to dose administration are possible. Appropriate drugs and medical equipment to treat acute anaphylactic reactions must be immediately available, and study personnel must be trained to recognize and treat anaphylaxis. The study site must have immediate access to emergency resuscitation teams and equipment in addition to the ability to admit subjects to an intensive care unit if necessary.

#### 5.1.5 Accountability and dispensation

Research pharmacy at each investigational site will be responsible for Durvalumab accountability and dispensation. The investigator's or site's designated investigational product manager is required to maintain accurate investigational product accountability records. Upon completion of the study, copies of investigational product accountability records will be returned to MedImmune.

## 5.1.6 Disposition of unused investigational study drug

All unused investigational product will be returned to a MedImmune authorized depot or disposed of upon authorization by MedImmune. The sites will account for all investigational study drug dispensed and also for appropriate destruction. Certificates of delivery and destruction must be signed.

Date 10/08/2018

#### 6. TREATMENT PLAN

## 6.1 Subject enrollment

Subjects with BCG refractory CIS urothelial carcinoma of the bladder as defined in inclusion criteria will be consented and screened.

Subjects who have completed 6 or more doses of Durvalumab and underwent month 6/week 26 bladder biopsy would be considered evaluable. Subjects who completed less than 6 doses of druvalumab will not be considered evaluable but will be followed until after the month 24 cystoscopic evaluation and biopsy. Subjects who withdrawn from the study prior to the month 6 cystoscopic evaluation and biopsy would be replaced to ensure a total of 34 evaluable subjects.

Subjects who are incorrectly enrolled but are not yet initiated on treatment should be withdrawn from the study.

## **6.2** Dosage and Administration

Durvalumab will be given every 4 weeks at 1500 mg IV for total of 12 months/13 doses (refer to Section 5.1.3 and 5.1.4 for the administration and monitoring of administration of durvalumab).

## 6.3 Durvalumab Dose Modification and Toxicity Management

For adverse events (AEs) that are considered at least partly due to administration of durvalumab, the following dose adjustment guidance may be applied:

- Treat each of the toxicities with maximum supportive care (including holding the agent suspected of causing the toxicity where required).
- If the symptoms promptly resolve with supportive care, consideration should be given to continuing the same dose of durvalumab along with appropriate continuing supportive care. If medically appropriate, dose modifications are permitted for durvalumab (see below).
- All dose modifications should be documented with clear reasoning and documentation of the approach taken.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

In addition, there are certain circumstances in which durvalumab should be permanently discontinued. These circumstances include but not limited to grade 3 toxicity at least possibly related to durvalumab; and prolonged grade 2 toxicity requiring dose delays for more than 2 weeks or requiring prolonged steroid use will discontinue durvalumab.

Following the first dose of durvalumab, subsequent administration of durvalumab can be modified based on toxicities observed (see Table 1, 2, and 3 in Appendix A). Dose reductions are not permitted.

Based on the mechanism of action of durvalumab leading to T-cell activation and proliferation, there is the possibility of observing immune related Adverse Events (irAEs) during the conduct of this study. Potential irAEs include immune-mediated enterocolitis, dermatitis, hepatitis, and endocrinopathies. Subjects should be monitored for signs and symptoms of irAEs. In the absence of an alternate etiology (e.g., infection or PD) signs or symptoms of enterocolitis, dermatitis, hepatitis, and endocrinopathy should be considered to be immune-related.

Dose modification recommendations and toxicity management guidelines for immune-mediated reactions, for infusion-related reactions, and for non-immune-mediated reactions are detailed in Tables 1, 2, and 3 respectively.

In addition, management guidelines for adverse events of special interest (AESIs) are detailed in Section 10.1.3. All toxicities will be graded according to NCI CTCAE V4.03.

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

# 7. RESTRICTIONS DURING THE STUDY AND CONCOMITANT TREATMENT(S)

## 7.1 Restrictions during the study

#### Contraception

Females of childbearing potential who are sexually active with a nonsterilized male partner must use 2 methods of effective contraception from screening, and must agree to continue using such precautions for at least 90 days following the last infusion of durvalumab; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.

- Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
- Subjects must use 2 acceptable methods of effective contraception as described in Table 4.
- Non-sterilized males who are sexually active with a female partner of childbearing potential must use 2 acceptable methods of effective contraception (see Table 4) from Day 1 and for 90 days after receipt of the final dose of investigational product.

Table 4. Effective methods of contraception (two methods must be used)

| Barrier Methods | Intrauterine Device Methods | Hormonal<br>Methods |
|---|---|---|
| Male condom plus spermicide | Copper T | Implants |
| Cap plus spermicide | Progesterone T <sup>a</sup> | Hormone shot or injection |
| Diaphragm plus spermicide | Levonorgestrel-releasing intrauterine system (e.g., Mirena®) <sup>a</sup> | Combined pill Minipill Patch |

a This is also considered a hormonal method.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

#### **Blood donation**

Subjects should not donate blood for at least 90 days following the last infusion of durvalumab.

## 7.2 Concomitant treatment(s)

## 7.2.1 Permitted concomitant medications

Investigators may prescribe concomitant medications or treatments (e.g., acetaminophen, diphenhydramine) deemed necessary to provide adequate prophylactic or supportive care except for those medications identified as "excluded" as listed in Section 7.2.2.

#### 7.2.2 Excluded Concomitant Medications

The following medications are considered exclusionary during the study.

- 1. Any investigational anticancer therapy
- 2. Any concurrent chemotherapy, radiotherapy (except palliative radiotherapy), immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable. <<NOTE: Local treatment of isolated lesions for palliative intent is acceptable (e.g., by local surgery or radiotherapy)>>
- 3. Immunosuppressive medications including, but not limited to systemic corticosteroids at doses not exceeding 10 mg/day of prednisone or equivalent, methotrexate, azathioprine, and TNF-α blockers. Use of immunosuppressive medications for the management of investigational product-related AEs or in subjects with contrast allergies is acceptable. In addition, use of inhaled and intranasal corticosteroids is permitted. <<A temporary period of steroids will be allowed for different indications, at the discretion of the principal investigator (e.g., chronic obstructive pulmonary disease, radiation, nausea, etc).>>
- 4. Live attenuated vaccines within 30 days of durvalumab dosing (ie, 30 days prior to the first dose, during treatment with durvalumab and for 30 days post discontinuation of durvalumab. Inactivated vaccines, such as the injectable influenza vaccine, are permitted.

Date 10/08/2018

| Table 5. Prohibited and Rescue Medications | |
|---|---|
| Rescue/supportive medication/class of drug: | Usage: |
| Concomitant medications or treatments (eg, acetaminophen or diphenhydramine) deemed necessary by the Investigator to provide adequate prophylactic or supportive care, except for those medications identified as "prohibited" as listed above | To be administered as prescribed by the Investigator |
| Best supportive care (including antibiotics, nutritional support, growth factor support, correction of metabolic disorders, optimal symptom control, and pain management [including palliative radiotherapy, etc]) | Should be used when necessary for all patients |

## 8. STUDY PROCEDURES

## 8.1 Schedule of study procedures

Before study entry, throughout the study, and following study drug discontinuation, various clinical and diagnostic laboratory evaluations are outlined. The purpose of obtaining these detailed measurements is to ensure adequate safety and tolerability assessments. Clinical evaluations and laboratory studies may be repeated more frequently if clinically indicated. The Schedules of Assessments during the screening and treatment period is provided following the Protocol Synopsis (note that these are the minimum requirements and the table will be adjusted according to each individual study).

#### 8.1.1 Screening Phase

Subjects with BCG refractory CIS urothelial bladder cancer will be consented and then screened for the study. Screening procedures will be performed up to 28 days before Day 1 Cycle 1, unless otherwise specified. All subjects must first read, understand, and sign the IRB/REB/IEC-approved ICF before any study-specific screening procedures are performed. After signing the ICF, completing all screening procedures, and being deemed eligible for entry, subjects will be enrolled in the study. Procedures that are performed prior to the signing of the ICF and are considered standard of care may be used as screening assessments if they fall within the 28-day screening window.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

The following procedures will be performed during the Screening Visit:

- Informed Consent
- Review of eligibility criteria
- Medical history and demographics
- Complete physical exam
- ECOG Performance Status
- Vitals signs, weight and height
- 12-lead ECG (in triplicate [2-5 minutes apart])
- Review of prior/concomitant medications
- CT urogram and chest X-ray to rule out metastasis
- Clinical laboratory tests for:
  - o Hematology (see Table 6)
  - o Clinical chemistry (see Table 7)
  - o TSH
  - o Coagulation (PT, PTT, INR)
  - o Creatinine Clearance
  - Serum pregnancy test (for women of childbearing potential only)
  - Hepatitis serologies
  - o Urinalysis (see Table 8)
  - Urine cytology with Urovysion FISH test

#### **8.1.2** Treatment Phase

Procedures to be conducted during the treatment phase of the study are presented in the Schedule of Assessments. Screening procedures performed within 72 hours of Cycle 1 Day 1 (C1D1) do not need to be repeated on C1D1.

#### **8.1.3** End of Treatment

End of treatment is defined as the last planned dosing visit within the 12-month dosing period. For subjects who discontinue durvalumab prior to 12 months, end of treatment is considered the last visit where the decision is made to discontinue treatment. All required procedures may be completed within  $\pm$  7 days of the end of treatment visit. <<Repeat disease assessment is not required if performed within 28 days prior to the end of treatment visit.>>

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

Assessments for subjects who have completed durvalumab treatment and achieved disease control, or have discontinued durvalumab due to toxicity in the absence of confirmed progressive disease are provided in APPENDIX C.

Assessments for subjects who have discontinued durvalumab treatment due to confirmed PD are presented in APPENDIX D.

## 8.2 Description of study procedures

# 8.2.1 Medical history and physical examination, electrocardiogram, weight and vital signs

Findings from medical history (obtained at screening) and physical examination shall be given a baseline grade according to the procedure for AEs. Increases in severity of pre-existing conditions during the study will be considered AEs, with resolution occurring when the grade returns to the pre-study grade or below.

Physical examinations will be performed on study days noted in the Schedule of Assessments.

A complete physical examination will be performed and will include an assessment of the following (as clinically indicated): general appearance, respiratory, cardiovascular, abdomen, skin, head and neck (including ears, eyes, nose and throat), lymph nodes, thyroid, musculo-skeletal (including spine and extremities), genital/rectal, and neurological systems and at screening only, height.

ECGs are required during screening as well as at any other time point when clinically indicated. ECGs recorded during the screening period will be obtained in triplicate (with 2-5 minute lag time between each). All 12-lead ECGs should be recorded while the subject is in the supine position for at least 5 minutes in each case.

Vital signs (temperature, blood pressure, pulse rate, and respiratory rate) will be measured on study days noted in the Schedule of Assessments. On durvalumab treatment days, vital signs will be measured within an hour prior to start of durvalumab administration, at 30 minutes during the infusion ( $\pm$  5 minutes), at the end of infusion ( $\pm$  5 minutes), and at 30 minutes ( $\pm$  5 minutes) and 60 minutes ( $\pm$  5 minutes) post-infusion. If the infusion takes longer than 60 minutes, then blood pressure and pulse measurements should follow the principles described here, or more frequently if clinically indicated. For subsequent doses, the 1-hour observation period will not be required unless a subject experiences an infusion-related reaction.

Date 10/08/2018

## 8.2.2 Clinical laboratory tests

The following clinical laboratory tests will be performed at each study site with reference range for each test provided (see the Schedule of Assessments, Appendix C and Appendix D for the timepoints of each test):

- Hematology (Table 6)
- Clinical Chemistry (Table 7)
- Coagulation parameters: Activated partial thromboplastin time and International normalised ratio to be assessed at baseline and as clinically indicated
- Urine analysis (Table 8)
- Urine cytology with Urovysion FISH test
- Thyroid Stimulating Hormone
  - o free T3 and free T4 only if TSH is abnormal
- Pregnancy test (female subjects of childbearing potential only)
  - o Urine human chorionic gonadotropin
  - o Serum beta-human chorionic gonadotropin (at screening only)
- Other laboratory tests
  - o Hepatitis B surface antigen, hepatitis C antibody
  - HIV antibody

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

#### **Table 6. Hematology Laboratory Tests**

Basophils Mean corpuscular volume

Eosinophils Monocytes
Hematocrit Neutrophils
Hemoglobin Platelet count

Lymphocytes Red blood cell count

Mean corpuscular hemoglobin Total white cell count

Mean corpuscular hemoglobin concentration

## Table7. Clinical chemistry (Serum or Plasma) Laboratory Tests

Albumin Glucose

Alkaline phosphatase Lactate dehydrogenase

Alanine aminotransferase Lipase

Amylase Magnesium
Aspartate aminotransferase Potassium
Bicarbonate Sodium

Calcium Total bilirubin<sup>a</sup>
Chloride Total protein

Creatinine Urea or blood urea nitrogen, depending on local practice

Gamma glutamyltransferase<sup>b</sup> Uric acid

## Table 8. Urinalysis Tests<sup>a</sup>

| Bilirubin | рН |
|-----------|-----------------------|
| Blood | Protein |
| Glucose | Specific gravity |
| Ketones | Colour and appearance |

<sup>&</sup>lt;sup>a</sup> If Total bilirubin is  $\ge 2xULN$  (and no evidence of Gilbert's syndrome) then fractionate into direct and indirect bilirubin

<sup>&</sup>lt;sup>b</sup> At baseline and as clinically indicated

<sup>a</sup> Microscopy should be used as appropriate to investigate white blood cells and use the high power field for red blood cells

## 8.3 Biological sampling procedures for PD-L1 testing

To ensure comparability of data across all studies of durvalumab, the Ventana SP263 assay will be used for testing PD-L1 expression. Testing should be restricted to the Ventana SP263 assay and should be performed in accordance with the package insert on the Ventana Benchmark platform (Ultra or XT).

The Ventana SP263 assay is fully analytically validated test characterized through to the completion of reader precision studies in the non-small cell lung cancer (NSCLC) and squamous cell carcinoma of the head & neck (SCCHN). For these tumors, the Ventana SP263 assay has a fully reproducibility data package supporting cut-off and scoring algorithm. Following completion of ATLANTIC and HAWK clinical trials, the assay will be associated with clinical utility. In other cancer types (bladder, pancreatic, gastric, hepatocellular, triple negative breast, ovarian, esophageal, nasopharyngeal, glioblastoma, soft tissue sarcoma, cholangiocarcinoma, small cell lung, melanoma and cervical HPV+ cancers), the Ventana SP263 assay has only limited clinical performance data.

#### Sample collection for PD-L1 testing

- The preferred tumor sample for the determination of a patient's PD-L1 status is the one taken following the completion of the most recent prior line of therapy. Samples taken at this time reflect the current PD-L1 status of the tumor and considered clinically most relevant.
- The preferred bladder biopsies or TURBT sample for PD-L1 testing was less than or
  equal to 90 days old. In cases where a sample of less than 90 days old was not
  available, patients were asked to undergo a new cystoscopic bladder biopsy and or
  TURBT.
- Samples should be evaluated for tumor cell quantity (i.e. >100 tumor cells) to allow for adequate PD-L1 immunohistochemistry analyses.
- When the collection of a new CIS sample with adequate tumor cell quantity is not clinically feasible, archival samples may be utilized provided the specimen it is not

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

older than 3 years of age. When archival samples are used to assess PD-L1 status, the age of the sample / date of collection should be captured.

• Samples submitted for PD-L1 testing should be formalin fixed and embedded in paraffin.

#### Sample data collection for PD-L1 testing

The following fields of data should be collected from the site/institution collecting and if, indicated shipping of the samples:

- Patient identifier (ecode or unique identifier)
- Specimen identifier (written on the specimen)
- Site identifier
- Specimen collection date
- Type of specimen submitted
- Quantity of specimen
- Date of sectioning
- Archival of fresh tumor
- Tumor type
- Primary tumor location
- Metastatic tumor location (if applicable)
- Fixative

## The following fields of data should be collected from PD-L1 testing laboratory:

- Are the negative and positive controls stained correctly
- Is the H&E material acceptable
- Is morphology acceptable
- Total percent positivity of PD-L1 in tumor cells
- PD-L1 status (positive, negative or NA) in tumor cells
- Total percent positivity of PD-L1 in infiltrating immune cells

The Ventana SP263 assay to measure PD-L1 in tumors is experimental. As with all tests, there is a chance of false positive (the test shows high PD-L1 when it is not there) or false negative (the test does not show PD-L1 when it is there) results may occur.

#### Sample processing and if indicated submission process for PD-L1 testing

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

#### Preparing Stored samples for testing

 Where samples already exist, they should be retrieved from the Bio-Bank storage location. These blocks should undergo quality review, prior to evaluation or shipment.
 Where it is not possible or indicated to ship the block to a testing laboratory, unstained slides should be prepared from the paraffin-embedded tumor sample block (described below) prior to evaluation or shipment.

#### Preparing newly acquired samples for PD-L1 testing

- If patients are undergoing a biopsy procedure that provides the option to submit newly acquired samples, this sample should be used to determine PD-L1 status. Where clinically acceptable, a minimum of 2 core biopsies should be collected and processed to FFPE in a single block. The provision of 2 cores is advised in order to provide sufficient tissue for PD-L1 assessment.
- Samples should be evaluated for tumor cell quantity (i.e. >100 tumor cells) and embedded in the same block.

#### Fixation of biopsy samples for PD-L1 testing

- Previously frozen tissue is not acceptable for processing to FFPE for PD-L1 testing. To fix newly acquired tissue, place immediately (within 30 min of excision) into an adequate volume of 10% v/v neutral buffered formalin (NBF). Samples should remain in fixative for 24 48 hours at room temperature.
- It is vital that there is an adequate volume of fixative relevant to the tissue (at least a 10 volume excess) and that large specimens (if any) are incised prior to fixation to promote efficient tissue preservation.

#### Embedding in paraffin for PD-L1 testing

- An overnight processing schedule into paraffin wax is recommended
- Below is the suggested routine overnight processing schedule:

#### Storage of tumor blocks for PD-L1 testing

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

• FFPE blocks should be stored at ambient temperature and protected from light until shipment by courier at ambient temperature. FFPE blocks are stable under these conditions for an indefinite period.

## Quality control of samples to be used for PD-L1 testing

- Tissue should be assessed by the site pathologist prior to PD-L1 testing.
- Each sample should be reviewed for:
  - Adequate fixation
  - Good preservation of morphology
  - Presence of tumor tissue
  - Histopathology consistent with indication
  - Greater than 100 tumor cells are required to determine PD-L1 status tumor cell content must be reviewed prior to testing in order for PD-L1 obtain a valid result.

## If indicated, shipping samples to a PD-L1 testing laboratory

• When submitting sample to for PD-L1 testing the recommendation is to ship the block in order for sectioning to occur at the laboratory. Blocks should be shipped containing enough material to be provided to allow a minimum of 5, and preferably 10, sections to be cut (each 4 micron thick) to be used for PD-L1 testing.

#### Sectioning instructions

- Where it is not possible or indicated to ship the block to laboratory for PD-L1 testing, unstained slides should be prepared from the paraffin-embedded tumor sample block as described below:
  - A minimum of 5-10 x 4 micron (μm) thick, unstained sections should be provided for PD-L1 testing
  - A new disposable microtome blade must be used for each block to prevent contamination between Slides are stable under these conditions for 6 months.
  - patient samples
  - Apply one section per slide to positively-charged Superfrost glass slides
  - The sections should be dried overnight between room temperature and 37°C. Do not dry sections at temperatures above 37°C.

Clinical Study Protocol
Drug Substance Durvalumab (Medi4736)
Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

Sections should be stored at ambient temperature and protected from light until use or shipment to testing lab by courier at ambient temperature. It is recommended that slides are cut freshly prior to PD-L1 testing and they are used within 90 days of being cut to obtain PD-L1 status.

## 9. DISEASE EVALUATION AND METHODS

The response to immunotherapy may differ from the typical responses observed with cytotoxic chemotherapy including the following (Wolchok et al 2009, Nishino et al 2013):

- Response to immunotherapy may be delayed
- Response to immunotherapy may occur after PD by conventional criteria
- The appearance of new lesions may not represent PD with immunotherapy
- SD while on immunotherapy may be durable and represent clinical benefit.

Based on the above-described unique response to immunotherapy, subjects with persistent CIS at the month 3 bladder biopsy will continue to receive Durvalumab until the month 6 bladder biopsy documented persistent CIS or progression to the muscle invasive stage. Durvalumab will be discontinued and subjects will be off study if invasive bladder cancer (T1 or above) is documented in any of the bladder biopsies. Due to the nature of CIS of bladder, RECIST 1.1 or irRECIST will not be applicable to response assessment.

#### 9.1.1 Pathological response

The absence of CIS of bladder on the mapping biopsies after pathological review would be considered complete response to treatment. Subjects who are withdrawn from durvalumab treatment for reasons other than confirmed progression to the muscle invasive stage will continue to have objective tumor assessments (see Appendix C).

## 9.1.2 Urine Cytology and UroVysion test

Positive urine cytology and or positive UroVysion test would indicate cancer either within or outside bladder (upper tract or prostatic uretheral). These data will be collected at baseline, month 6, and 24. Only pathological response will be used to assess the primary and secondary objectives.

Date 10/08/2018

## 9.1.3 Compare the tumor mutation burden and alterations in DNA repair genes in the pre and post Durvalumab urothelial bladder cancer samples

This will be performed on the TEMPUS xT gene panel, which detects single nucleotide variants, indels, and copy number variant in 595 genes with tumor DNA sequencing. Microsatellite instability status and tumor mutation burden will be reported as well.

## 10. ASSESSMENT OF SAFETY

The Principal Investigator is responsible for ensuring that all staff involved in the study is familiar with the content of this section.

## 10.1 Safety Parameters

#### 10.1.1 Definition of adverse events

The International Conference on Harmonization (ICH) Guideline for Good Clinical Practice (GCP) E6 (R1) defines an AE as:

Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

An AE includes but is not limited to any clinically significant worsening of a subject's pre-existing condition. An abnormal laboratory finding (including ECG finding) that requires an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation, should be reported as an AE.

Adverse events may be treatment emergent (ie, occurring after initial receipt of investigational product) or nontreatment emergent. A nontreatment-emergent AE is any new sign or symptom, disease, or other untoward medical event that begins after written informed consent has been obtained but before the subject has received investigational product.

Elective treatment or surgery or preplanned treatment or surgery (that was scheduled prior to the subject being enrolled into the study) for a documented pre-existing condition, that did not worsen from baseline, is not considered an AE (serious or nonserious). An untoward medical

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

event occurring during the prescheduled elective procedure or routinely scheduled treatment should be recorded as an AE or SAE.

The term AE is used to include both serious and non-serious AEs.

#### 10.1.2 Definition of serious adverse events

A serious adverse event is an AE occurring during any study phase (i.e., screening, run-in, treatment, wash-out, follow-up), at any dose of the study drugs that fulfils one or more of the following criteria:

Results in death

Is immediately life-threatening

Requires in-patient hospitalization or prolongation of existing hospitalization

Results in persistent or significant disability, incapacity, or substantial disruption of the ability to conduct normal life functions

Is a congenital abnormality or birth defect in offspring of the subject

Is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.

Medical or scientific judgment should be exercised in deciding whether expedited reporting is appropriate in this situation. Examples of medically important events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalizations; or development of drug dependency or drug abuse.

The causality of SAEs (their relationship to all study treatment/procedures) will be assessed by the investigator(s) and communicated to AstraZeneca.

## 10.1.3 Definition of adverse events of special interest (AESI)

An adverse event of special interest (AESI) is one of scientific and medical interest specific to understanding of durvalumab and may require close monitoring and rapid communication by the investigator to the sponsor. An AESI may be serious or non-serious. The rapid reporting of AESIs allows ongoing surveillance of these events in order to characterize and understand them in association with the use of durvalumab.

AESIs for durvalumab include but are not limited to events with a potential inflammatory or immune-mediated mechanism and which may require more frequent monitoring and/or interventions such as steroids, immunosuppressants and/or hormone replacement therapy.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

These AESIs are being closely monitored in clinical studies with durvalumab monotherapy and combination therapy. An immune-related adverse event (irAE) is defined as an adverse event that is associated with drug exposure and is consistent with an immune-mediated mechanism of action and where there is no clear alternate aetiology. Serologic, immunologic, and histologic (biopsy) data, as appropriate, should be used to support an irAE diagnosis. Appropriate efforts should be made to rule out neoplastic, infectious, metabolic, toxin, or other etiologic causes of the irAE.

If the Investigator has any questions in regards to an adverse event (AE) being an irAE, the Investigator should promptly contact the Study Physician.

AESIs observed with durvalumab include:

- Colitis
- Pneumonitis
- ALT/AST increases / hepatitis / hepatotoxicity
- Neuropathy / neuromuscular toxicity (i.e. events of encephalitis, peripheral motor and sensory neuropathies, Guillain-Barré, and myasthenia gravis)
- Endocrinopathy (i.e. events of hypophysitis, adrenal insufficiency, and hyper- and hypothyroidism)
- Dermatitis
- Nephritis
- Pancreatitis (or labs suggestive of pancreatitis increased serum lipase, increased serum amylase)

Further information on these risks (e.g. presenting symptoms) can be found in the current version of the durvalumab Investigator Brochure.

#### 10.1.4 Pneumonitis

Adverse events of pneumonitis are of interest for AstraZeneca/Medimmune, as pneumonitis, interstitial lung disease (ILD) has been reported with anti-PD-1 MAbs (Topalian et al, NEJM 2012). Initial work-up should include high-resolution CT scan, ruling out infection, and pulse oximetry. Pulmonary consultation is highly recommended.

Guidelines for the management of subjects with immune-mediated events including pneumonitis are outlined in Section 6.6.1.

#### **10.1.5** Hypersensitivity Reactions

Hypersensitivity reactions as well as infusion-related reactions have been reported with anti-PD-L1 and anti-PD-1 therapy (Brahmer et al 2012). As with the administration of any foreign protein and/or other biologic agents, reactions following the infusion of MAbs can be caused by various mechanisms, including acute anaphylactic (immunoglobulin E-mediated) and

anaphylactoid reactions against the MAb, and serum sickness. Acute allergic reactions may occur, may be severe, and may result in death. Acute allergic reactions may include hypotension, dyspnea, cyanosis, respiratory failure, urticaria, pruritus, angioedema, hypotonia, arthralgia, bronchospasm, wheeze, cough, dizziness, fatigue, headache, hypertension, myalgia, vomiting and unresponsiveness.

Guidelines for management of subjects with hypersensitivity (including anaphylactic reaction) and infusion-related reactions are outlined in Section 6.6.1.

#### 10.1.6 Hepatic function abnormalities (hepatotoxicity)

Increased transaminases have been reported during treatment with anti-PD-L1/anti-PD-1 antibodies (Brahmer et al 2012). Inflammatory hepatitis has been reported in 3% to 9% of subjects treated with anti-CTLA-4 monoclonal antibodies (e.g., ipilimumab). The clinical manifestations of ipilimumab-treated subjects included general weakness, fatigue, nausea and/or mild fever and increased liver function tests such as AST, ALT, alkaline phosphatase, and/or total bilirubin.

Hepatic function abnormality is defined as any increase in ALT or AST to greater than  $3 \times \text{ULN}$  and concurrent increase in total bilirubin to be greater than  $2 \times \text{ULN}$ . Concurrent findings are those that derive from a single blood draw or from separate blood draws taken within 8 days of each other. Follow-up investigations and inquiries will be initiated promptly by the investigational site to determine whether the findings are reproducible and/or whether there is objective evidence that clearly supports causation by a disease (e.g., cholelithiasis and bile duct obstruction with distended gallbladder) or an agent other than the investigational product. Guidelines for management of subjects with hepatic function abnormality are outlined in Table 1.

Cases where a subject shows an AST or ALT  $\ge 3x$ ULN or total bilirubin  $\ge 2x$ ULN may need to be reported as SAEs, These cases should be reported as SAEs if, after evaluation they meet the criteria for a Hy's Law case or if any of the individual liver test parameters fulfill any of the SAE criteria.

#### 10.1.7 Gastrointestinal disorders

Guidelines on management of diarrhea and colitis in patients receiving durvalumab are provided in Table 1.

#### 10.1.8 Endocrine disorders

Immune-mediated endocrinopathies include hypophysitis, adrenal insufficiency, and hyperand hypothyroidism. Guidelines for the management of patients with immune-mediated endocrine events are provided in Table 1.

#### 10.1.9 Pancreatic disorders

Immune-mediated pancreatitis includes autoimmune pancreatitis, and lipase and amylase elevation. Guidelines for the management of patients with immune-mediated pancreatic disorders are provided in Table 1.

#### 10.1.10 Neurotoxicity

Immune-mediated nervous system events include encephalitis, peripheral motor and sensory neuropathies, Guillain-Barré, and myasthenia gravis. Guidelines for the management of patients with immune-mediated neurotoxic events are provided in Table 1.

#### 10.1.11 Nephritis

Consult with Nephrologist. Monitor for signs and symptoms that may be related to changes in renal function (e.g. routine urinalysis, elevated serum BUN and creatinine, decreased creatinine clearance, electrolyte imbalance, decrease in urine output, proteinuria, etc)

Patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression, infections etc.)

Steroids should be considered in the absence of clear alternative etiology even for low grade events (Grade 2), in order to prevent potential progression to higher grade event. Guidelines for the management of patients with immune-mediated neurotoxic events are provided in Table 1.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

#### Criteria for Hy's Law (FDA Guidance 2009)

- The drug causes hepatocellular injury, generally shown by a higher incidence of 3-fold or greater elevations above the ULN of ALT or AST than the (non-hepatotoxic) control drug or placebo
- Among trial subjects showing such aminotransferase elevations, often with aminotransferases much greater than 3 x ULN, one or more also show elevation of serum total bilirubin to >2 x ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)
- No other reason can be found to explain the combination of increased aminotransferases and total bilirubin, such as viral hepatitis A, B, or C; pre-existing or acute liver disease; or another drug capable of causing the observed injury.

## 10.2 Assessment of safety parameters

## 10.2.1 Assessment of severity

Assessment of severity is one of the responsibilities of the investigator in the evaluation of AEs and SAEs. Severity will be graded according to the NCI CTCAE v4.03. The determination of severity for all other events not listed in the CTCAE should be made by the investigator based upon medical judgment and the severity categories of Grade 1 to 5 as defined below.

Grade 1 (mild) An event that is usually transient and may require only minimal

treatment or therapeutic intervention. The event does not generally

interfere with usual activities of daily living.

Grade 2 (moderate) An event that is usually alleviated with additional specific therapeutic

intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm

to the subject.

Grade 3 (severe) An event that requires intensive therapeutic intervention. The event

interrupts usual activities of daily living, or significantly affects the

clinical status of the subject.

Grade 4 (life threatening) An event, and/or its immediate sequelae, that is associated with

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

an imminent risk of death or with physical or mental disabilities that affect or limit the ability of the subject to perform activities of daily living (eating, ambulation, toileting, etc).

Grade 5 (fatal) Death (loss of life) as a result of an event.

It is important to distinguish between serious criteria and severity of an AE. Severity is a measure of intensity whereas seriousness is defined by the criteria in Section 10.1.2. A Grade 3 AE need not necessarily be considered an SAE. For example, a Grade 3 headache that persists for several hours may not meet the regulatory definition of an SAE and would be considered a nonserious event, whereas a Grade 2 seizure resulting in a hospital admission would be considered an SAE.

#### 10.2.2 Assessment of relationship

Assessment of relationship between AEs and Durvalumab will be performed by the treating physician/investigator at the time of each clinic visit. Such assessment will be based on investigators clinical judgment and the known AEs of Druvalumab.

## 10.3 Recording of adverse events and serious adverse events

Adverse events will be recorded using a recognized medical term or diagnosis that accurately reflects the event and captured in OnCore. Adverse events will be assessed by the investigator for severity, relationship to the investigational product, possible etiologies, and whether the event meets criteria of an SAE and therefore requires immediate notification to AstraZeneca/MedImmune Patient Safety.

The following variables will be collected for each AE:

- AE (verbatim)
- The date when the AE started and stopped
- Changes in NCI CTCAE grade and the maximum CTC grade attained
- Whether the AE is serious or not
- Investigator causality rating against durvalumab
- Action taken with regard to durvalumab /comparator/combination agent
- Outcome

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

In addition, the following variables will be collected for SAEs as applicable:

- Date AE met criteria for serious AE
- Date Investigator became aware of serious AE
- AE is serious due to <<criteria>>
- Date of hospitalization
- Date of discharge
- Probable cause of death
- Date of death
- Autopsy performed
- Description of AE
- Causality assessment in relation to Study procedure(s)

Events, which are unequivocally due to disease progression, should not be reported as an AE during the study. Disease progression can be considered as a worsening of a patient's condition attributable to the disease for which the investigational product is being studied. It may be an increase in the severity of the disease under study and/or increases in the symptoms of the disease. The development of new metastasis of the primary cancer under study should be considered as disease progression and not an AE.

## 10.3.1 Study recording period and follow-up for adverse events and serious adverse events

Adverse events and serious adverse events will be recorded from time of signature of informed consent, throughout the treatment period and including the follow-up period (90 days after the last dose of durvalumab)

During the course of the study all AEs and SAEs should be proactively followed up for each subject. Every effort should be made to obtain a resolution for all events, even if the events continue after discontinuation/study completion.

If a subject discontinues from treatment for reasons other than disease progression, and therefore continues to have tumor assessments, drug or procedure-related SAEs must be captured until the patient is considered to have confirmed PD and will have no further tumor assessments.

The investigator is responsible for following all SAEs until resolution, until the subject returns to baseline status, or until the condition has stabilized with the expectation that it will remain chronic, even if this extends beyond study participation.

#### Follow-up of unresolved adverse events

Any AEs that are unresolved at the subject's last visit in the study are followed up by the investigator for as long as medically indicated, but without further recording in the eCRF. After 90 days, only subjects with ongoing investigational product-related SAEs will continue to be followed for safety.

AstraZeneca/MedImmune retains the right to request additional information for any subject with ongoing AE(s)/SAE(s) at the end of the study, if judged necessary.

#### Post study events

After the subject has been permanently withdrawn from the study, there is no obligation for the investigator to actively report information on new AE or SAEs occurring in former study subjects after the 90-day safety follow-up period for patients treated with durvalumab. However, if an investigator learns of any SAEs, including death, at any time after the subject has been permanently withdrawn from study, and he/she considers there is a reasonable possibility that the event is related to study treatment, the investigator should notify the study sponsor and AstraZeneca/MedImmune Drug Safety.

#### **10.3.2** Reporting of serious adverse events

Information about all serious adverse events will be collected and recorded. All SAEs will be reported, whether or not considered causally related to the investigational product, or to the study procedure(s). The reporting period for SAEs is the period immediately following the time that written informed consent is obtained through 90 days after the last dose of durvalumab or until the initiation of alternative anticancer therapy. To ensure patient safety, each serious adverse event must be reported to the PI and to the sponsor expeditiously. Moffitt Cancer Center and all participating sites will report SAEs by completing an SAE report in OnCore, the electronic data capture system. The SAE must be reported by email (affiliate.research@moffitt.org) to the External Site Coordination (ESC) office within 2 working days. If applicable, the site should also follow protocol guidelines for additional reporting to government agencies.

The investigator and Sponsor are responsible for informing the Regulatory Authority of the SAE as per local requirements.

The investigator and/or sponsor must inform the FDA, via a MedWatch/AdEERs form, of any serious or unexpected adverse events that occur in accordance with the reporting obligations of 21 CFR 312.32, and will concurrently forward all such reports to AstraZeneca. A copy of the MedWatch/AdEERs report must be faxed to AstraZeneca at the time the event is reported

to the FDA. It is the responsibility of the sponsor to compile all necessary information and ensure that the FDA receives a report <u>according to the FDA reporting requirement timelines</u> and to ensure that these reports are also submitted to AstraZeneca at the same time.

\* A cover page should accompany the MedWatch/AdEERs form indicating the following:

"Notification from an Investigator Sponsored Study"

The investigator IND number assigned by the FDA

The investigator's name and address

The trial name/title and AstraZeneca ISS reference number (ESR-##-#####)

- \* Sponsor must also indicate, either in the SAE report or the cover page, the *causality* of events *in relation to all study medications* and if the SAE is *related to disease progression*, as determined by the principal investigator.
- \* Send SAE report and accompanying cover page by way of email to AstraZeneca's designated mailbox: AEMailboxClinicalTrialTCS@astrazeneca.com

If a non-serious AE becomes serious, this and other relevant follow-up information must also be provided to AstraZeneca and the FDA.

Serious adverse events that do not require expedited reporting to the FDA still need to be reported to AstraZeneca preferably using the MedDRA coding language for serious adverse events. This information should be reported on a monthly basis and under no circumstance less frequently than quarterly.

#### 10.3.3 Reporting of deaths

All deaths that occur during the study, or within the protocol-defined 90-day post-last dose of durvalumab safety follow-up period must be reported as follows:

Death that is clearly the result of disease progression should be documented but should not be reported as an SAE.

Where death is not due (or not clearly due) to progression of the disease under study, the AE causing the death must be reported to as a SAE within **24 hours** (see Section 10.3.2 for further details). The report should contain a comment regarding the co-involvement of progression of disease, if appropriate, and should assign main and contributory causes of death.

Deaths with an unknown cause should always be reported as a SAE.

Date 10/08/2018

Deaths that occur following the protocol-defined 90-day post-last-dose of durvalumab safety follow-up period will be documented <<as events for survival analysis>>, but will not be reported as an SAE.

## 10.3.4 Other events requiring reporting

#### 10.3.5 Overdose

An overdose is defined as a subject receiving a dose of durvalumab in excess of that specified in the Investigator's Brochure, unless otherwise specified in this protocol.

Any overdose of a study subject with durvalumab, with or without associated AEs/SAEs, is required to be reported within 24 hours of knowledge of the event to the sponsor and AstraZeneca/MedImmune Patient Safety or designee using the designated Safety e-mailbox (see Section 10.3.2 for contact information). The following information should be provided in the event of an Overdose (Overdose Report Form can be provided upon request):

- Details of the Patient who was dispensed study medication (Randomization code)
- Details of the Patient who took the overdose (demographic information, was patient a study participant?)
- Details of the drug overdose (total daily dose, route, formulation, Overdose start and stop dates)
- Was the overdose accidental or intentional?
- Was the overdose associated with an adverse event (serious or non-serious)
- Provide an Adverse Event description (use same wording as in CRF). Provide start and stop dates of the event, or indicate if the event is ongoing.
- Provide Investigator's signature and date.

If the overdose results in an AE, the AE must also be recorded as an AE (see Section 10.3). Overdose does not automatically make an AE serious, but if the consequences of the overdose are serious, for example death or hospitalization, the event is serious and must be recorded and reported as an SAE (see Section 10.1.2 and Section 10.3.2). There is currently no specific treatment in the event of an overdose of durvalumab.

The investigator will use clinical judgment to treat any overdose.

#### 10.3.6 Hepatic function abnormality

Hepatic function abnormality (as defined in Section 10.1.3.3) in a study subject, with or without associated clinical manifestations, is required to be reported as "hepatic function abnormal" within 24 hours of knowledge of the event to the sponsor and

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

AstraZeneca/MedImmune Patient Safety using the designated Safety e-mailbox (see Section 10.3.2 for contact information), unless a definitive underlying diagnosis for the abnormality (e.g., cholelithiasis or bile duct obstruction) that is unrelated to investigational product has been confirmed.

- If the definitive underlying diagnosis for the abnormality has been established and is unrelated to investigational product, the decision to continue dosing of the study subject will be based on the clinical judgment of the investigator.
- If no definitive underlying diagnosis for the abnormality is established, dosing of the study subject must be interrupted immediately. Follow-up investigations and inquiries must be initiated by the investigational site without delay.

Each reported event of hepatic function abnormality will be followed by the investigator and evaluated by the sponsor and AstraZeneca/MedImmune.

## 10.3.7 Pregnancy

#### 10.3.8 Maternal exposure

If a patient becomes pregnant during the course of the study, the IPs should be discontinued immediately.

Pregnancy itself is not regarded as an AE unless there is a suspicion that the IP under study may have interfered with the effectiveness of a contraceptive medication. Congenital abnormalities or birth defects and spontaneous miscarriages should be reported and handled as SAEs. Elective abortions without complications should not be handled as AEs. The outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth, or congenital abnormality) should be followed up and documented even if the patient was discontinued from the study.

If any pregnancy occurs in the course of the study, then the Investigator or other site personnel should inform the appropriate AstraZeneca representatives within 1 day, ie, immediately, but **no later than 24 hours** of when he or she becomes aware of it.

The designated AstraZeneca representative will work with the Investigator to ensure that all relevant information is provided to the AstraZeneca Patient Safety data entry site within 1 to 5 calendar days for SAEs and within 30 days for all other pregnancies.

The same timelines apply when outcome information is available.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

#### 10.3.9 Paternal exposure

Male patients should refrain from fathering a child or donating sperm during the study and for 90 days after the last dose of durvalumab monotherapy.

Pregnancy of the patient's partner is not considered to be an AE. However, the outcome of all pregnancies (spontaneous miscarriage, elective termination, ectopic pregnancy, normal birth, or congenital abnormality) occurring from the date of the first dose until 90 days after the last dose should, if possible, be followed up and documented.

Where a report of pregnancy is received, prior to obtaining information about the pregnancy, the Investigator must obtain the consent of the patient's partner. Therefore, the local study team should adopt the generic ICF template in line with local procedures and submit it to the relevant Institutional Review Boards (IRBs) prior to use.

# 11. STATISTICAL METHODS AND SAMPLE SIZE DETERMINATION

## 11.1 Description of analysis sets

#### 11.1.1 Safety analysis set

Subjects who have received at least one dose of Durvalumab will be included in the Safety Analysis Set

#### 11.1.2 Efficacy analysis set

Subjects who have completed at least 6 treatments of every 4 week Durvalumab IV infusions and underwent the month 6 mapping biopsy will be included in the efficacy analysis set. Intention to treat analysis will be performed on all subjects who have completed at least one dose of Durvalumab and underwent the month 6 mapping biopsy.
# 11.2 Methods of statistical analyses

The null hypothesis that the 18% historical complete response rate at month 6 will be tested against a one-sided alternative of 40% or higher complete response rate with Durvalumab at month 6 in BCG refectory CIS of bladder. We use a Simon's two-stage design (Simon, 1989) based on the optimal two-stage designs and admissible designs (Jung et al. 2004) for Phase II single arm clinical trials.

In the first stage of this study plan, 13 patients will be accrued. If there are 3 or fewer responses in these 13 patients, the study will be stopped. Otherwise, 21 additional patients will be accrued for a total of 34. The null hypothesis will be rejected if 9 or more responses are observed in 34 patients. In summary 34 is the total number of subjects required, 13 is the number of subjects accrued during stage 1, if 3 or fewer responses are observed during stage 1, the trial is stopped early for futility, and, if 9 or fewer responses are observed by the end of stage two, then no further investigation of the drug is warranted. This design yields a one-sided type I error rate of 0.047 and power of 80% when the true response rate is 40%.

The primary analysis will be performed for the (complete) response rate based on month 6 mapping biopsy. We will use an exact probability method such as Chi-square and binomial tests.

| n | n <sub>1</sub> | <i>r</i> <sub>1</sub> | <b>r</b> 2 | Type 1 Error | Power | EN <sub>0</sub> | Probability of early stopping | Interval for w | Comment |
|---|---|---|---|---|---|---|---|---|---|
| 34 | 13 | 3 | 9 | 0.0473 | 0.8031 | 17.1 | 0.8061 | [0,0.1243] | Optimal |

EN0 is the expected sample size for the trial when response rate is p0 Interval for w is the set of values w such that the design minimizes w \* 21 + (1 - w) \* EN0

# 11.2.1 Safety Analyses

Descriptive statistics will be applied to safety analysis

## 11.2.2 Efficacy Analyses

Descriptive statistics will be applied to Efficacy analyses/pathological response rates at month 6 and 24.

## 11.2. 3 Exploratory Analysis

Due to the small sample size, descriptive statistics will be applied to assess putative associations between pathological response rates at month 6 and 24 and PD-L1 IHC positivity; between pathological response rates and chromosomal abnormalities observed in the Urovysion test. PD-L1 IHC on formalin-fixed paraffin-embedded tumor blocks will be performed by AstraZeneca. Urine Urovysion test is a standard of care test and will be performed at Moffitt Cancer Center.

## 11.2.3 Interim analyses

Interim analysis of this study will be performed when 13 patients have been enrolled and completed the protocol required month 6 biopsy. If there are 3 or fewer responses in these 13 patients, the study will be stopped. Otherwise, the study will be continued and 21 additional patients will be accrued for a total of 34.

# 11.3 Determination of sample size

The required total number of subjects is 34. 13 is the number of subjects accrued during stage 1. If 3 or fewer responses are observed during stage 1, the trial is stopped early for futility. If 9 or fewer responses of total 34 patients are observed by the end of stage two, then no further investigation of the drug is warranted. This design yields a one-sided type I error rate of 0.047 and power of 80% when the true response rate is 40% based on Simon's optimal two-stage design.

# 12. ETHICAL AND REGULATORY REQUIREMENTS

# 12.1 Ethical conduct of the study

The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, and applicable regulatory requirements Subject data protection.

Date 10/08/2018

# 12.2 Ethics and regulatory review

Institution's scientific review committee (SRC) conducts a formal internal peer review of all clinical protocols and general scientific oversight of interventional clinical research. Protocols are reviewed for scientific merit, adequate study design, safety, availability of targeted study population, and feasibility of timely completion of all proposed research projects to be conducted by its assigned programs at the Cancer Center. The SRC is responsible for evaluating the risk/benefit assessment and corresponding data and safety monitoring plan as part of the scientific review and approval process.

An IRB should approve the final study protocol, including the final version of the ICF and any other written information and/or materials to be provided to the subjects. The investigator will ensure the distribution of these documents to the applicable IRB, and to the study site staff. The review of this protocol by the IRB and the performance of all aspects of the study, including the methods used for obtaining informed consent, must also be in accordance with principles enunciated in the declaration, as well as ICH Guidelines, Title 21 of the Code of Federal Regulations (CFR), Part 50 Protection of Human Subjects and Part 56 Institutional Review Boards.

The approval for both the protocol and informed consent must specify the date of approval, protocol number and version, or amendment number. Principal investigator at each site is responsible for providing the IRB with reports of any serious and unexpected adverse drug reactions from any other study conducted with Durvalumab.

## 12.3 Informed consent

The Principal Investigator(s) at each center will:

- Ensure each subject is given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study
- Ensure each subject is notified that they are free to discontinue from the study at any time
- Ensure that each subject is given the opportunity to ask questions and allowed time to consider the information provided
- Ensure each subject provides signed and dated informed consent before conducting any procedure specifically for the study
- Ensure the original, signed ICF(s) is/are stored in the Investigator's Study File

- Ensure a copy of the signed ICF is given to the subject
- Ensure that any incentives for subjects who participate in the study as well as any provisions for subjects harmed as a consequence of study participation are described in the ICF that is approved by an IRB

# 12.4 Changes to the protocol and informed consent form

If there are any substantial changes to the study protocol, then these changes will be documented in a study protocol amendment and where required in a new version of the study protocol. The amendment is to be approved by the relevant IRB/IEC and if applicable, also the SRC, before implementation.

# 12.5 Audits and inspections

Authorized representatives of Moffitt cancer center, a regulatory authority, or an IRB may perform audits or inspections at the center, including source data verification. The purpose of an audit or inspection is to systematically and independently examine all study-related activities and documents, to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, Good Clinical Practice, guidelines of the ICH, and any applicable regulatory requirements.

## 13. STUDY MANAGEMENT

# 13.1 Training of study site personnel

Before the first subject is entered into the study, principle investigators at each site will review and discuss the requirements of the clinical study protocol and related documents with the investigational staff and also train them in any study-specific procedures and system(s) utilized. The principal investigator will ensure that appropriate training relevant to the study is given to all of these staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

The principal investigator will maintain a record of all individuals involved in the study

# **Monitoring of the study**

The protocol monitoring committee (PMC) at Moffitt cancer center meets once a month. The PMC reviews and evaluates safety and/or efficacy data for all physician authored clinical intervention trials. The PMC ensures the safety of patients and the validity and integrity of data. PMC reviews SAEs, deviations, Interim analysis, interim and final reports from the external Data Monitoring Committee (DMC) as well as audits both internally and externally.

The PMC can make the following determinations, Accepted, Acceptable with Corrective Action and Tabled.

# 13.3 Study timetable and end of study

We anticipate having the study open for enrollment at Moffitt in February 2017 and have the study open at additional sites before December 2018. We plan to complete enrollment of the first 13 pilot subjects in 6 months. If more than 3 of the first13 subjects responded to therapy, the study will proceed with enrolling total of 34 subjects. We anticipate enrolling the last subject in December 2019 and end the study in December 2021.

# 13.4 Affiliate Sites Required Documentation

Before the study can be initiated at any site, the site will be required to provide regulatory documentation to the External Site Coordination (ESC) office at Moffitt Cancer Center. Sites must provide a copy of their informed consent to the ESC office for review and approval prior to submission of any documents to the site's IRB. Any changes requested by the site's IRB must be provided to the ESC staff for review and approval prior to resubmission to the IRB.

The ESC office must receive the following trial specific documents either by hardcopy, fax, or email before a site can be activated for any trial:

- 1. IRB Approval Letter that includes the protocol version and date
- 2. FDA Related Forms 1572/1571/310 as appropriate
- 3. Signed Protocol Title Page
- 4. IRB Approved Consent Form
- 5. Site Delegation of Authority Log
- 6. Signed Financial Interest Disclosure Forms (principal and sub investigators)
- 7. Updated Investigator/Personnel documents (CVs, licenses, GCP and HSP training certificates, etc.) as needed
- 8. Updated Laboratory Documents (certifications, normal ranges, etc.) as needed
- 9. Signed protocol specific Task Order

A study initiation teleconference will be held prior to the start of any study related activity at the site. Attendance is required for:

- The site PI and appropriate research staff
- Moffitt PI and ESC research coordinator

The requirements of the protocol and all associated procedures and processes will be reviewed and agreed upon prior to the activation of the study. The ESC utilizes the EDC system, OnCore. OnCore training will be scheduled, if indicated, with the appropriate staff from the site.

## 14. DATA MANAGEMENT

The Principal Investigator and the Clinical Research Coordinator assigned to the case will be primarily responsible for maintaining all study related documents including the clinical research forms. Oncore is Moffitt's clinical trial database of record for all CRF entries and will be verified with source documentation. The review of medical records within PowerChart will be done in a manner to assure that patient confidentiality is maintained. Regulatory documents and case report forms will be reviewed routinely for accuracy, completeness and source verification of data entry, validation of appropriate informed consent process, adherence to study procedures, and reporting of SAEs and protocol deviations according to Moffitt's Monitoring Policies.

## 14.1 Data Management and Monitoring/Auditing

Data will be captured in OnCore, Moffitt's Clinical Trials Database. Regulatory documents and case report forms will be monitored internally according to Moffitt Cancer Center Monitoring Policies. Monitoring will be performed regularly to verify data is accurate, complete, and verifiable from source documents; and the conduct of the trial is in compliance with the currently approved protocol/amendments, Good Clinical Practice (GCP), and applicable regulatory requirements.

To obtain access to OnCore, the External Site Coordination (ESC) office Coordinator will supply forms required to be completed by the site staff. Once the completed forms are received, the site coordinator will receive DUO access, logon/password, and information on how to access OnCore. The ESC office will provide OnCore training to the site once initial access is granted and on an ongoing basis, as needed.

# 14.2 Study governance and oversight

The safety of all AstraZeneca clinical studies is closely monitored on an ongoing basis by AstraZeneca representatives in consultation with Patient Safety. Issues identified will be addressed; for instance, this could involve amendments to the study protocol and letters to Investigators.

Date 10/08/2018

## 15. INVESTIGATIONAL PRODUCT AND OTHER TREATMENTS

# 15.1 Identity of investigational product(s)

| Table 1. List of investigational products for this study | | |
|---|---|---|
| Investigational product Dosage form and strength Manufacturer | | |
| Durvalumab | 1500 mg, solution, IV | MedImmune |

## 16. LIST OF REFERENCES

Andorsky DJ, Yamada RE, Said J, Pinkus GS, Betting DJ, and Timmerman JM. Programmed death ligand 1 is expressed by non-hodgkin lymphomas and inhibits the activity of tumorassociated T cells. Clin Cancer Res. 2011. 17(13):4232-4244.

Bellati F, Napoletano C, Ruscito I, et al: Past, present and future strategies of immunotherapy in gynecological malignancies. Curr Mol Med 2013; 13:648-69.

Bookman MA, Brady MF, McGuire WP, et al: Evaluation of new platinum-based treatment regimens in advanced-stage ovarian cancer: a Phase III Trial of the Gynecologic Cancer Intergroup. J Clin Oncol 2009; 27:1419-25.

Brahmer JR, Tykodi SS, Chow LQM, Hwu WJ, Topalian SL, Hwu P, et al. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65.

Brusa D, Serra S, Coscia M, Rossi D, D'Arena G, Laurenti L, et al. The PD-1/PD-L1 axis contributes to T-cell dysfunction in chronic lymphocytic leukemia. Haematologica. 2013 Jun; 98(6):953-963.

Burger RA, Brady MF, Bookman MA, et al: Incorporation of bevacizumab in the primary treatment of ovarian cancer. The New England journal of medicine 2011; 365:2473-83.

Callahan MK and Wolchok JD. CTLA-4 and PD-1 blocking antibodies in cancer immunotherapy. J Leukoc Biol. 2013; 94(1):41-53.

Date 10/08/2018

Chow et al. Exploring novel immune-related toxicities and endpoints with immune-checkpoint inhibitors in non-small cell lung cancer. Am Soc Clin Oncol Educ Book. 2013

Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16(1):31-41.

Coleman RL, Monk BJ, Sood AK, et al: Latest research and treatment of advanced-stage epithelial ovarian cancer. Nature Reviews Clinical Oncology 2013; 10:211-224.

Dinney CP, Greenberg RE, Steinberg GD. Intravesical valrubicin in patients with bladder carcinoma in situ and contraindication to or failure after bacillus Calmette-Guérin. Urol Oncol. 2013;31(8):1635-42

Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, et al. New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45:228-47.

European Medicines Agency's "Guideline on the evaluation of anti-cancer medicinal products in man" (EMA/CHMP/205/95/Rev.4)

Fagotti A, Ferrandina G, Fanfani F, et al: A laparoscopy-based score to predict surgical outcome in patients with advanced ovarian carcinoma: a pilot study. Ann Surg Oncol 2006; 13:1156-61.

Fellman, B. M. Stata command for calculating adverse event and efficacy stopping boundaries for phase II single-arm trials. *Stata Journal*. 2014; 14(2):407-417.

Food and Drug Administration Guidance for Industry (issued July 2009) 'Drug-induced liver injury: Premarketing clinical evaluation'. Available from URL: http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM174090.pdf. Accessed 10 December 2013.

Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, et al. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Nat Acad Sci U S A. 2007;104(9):3360-5.

Hamid et al. Safety and tumor responses with lambrolizumab (anti-PD-1) in melanoma.  $\underline{N}$  Engl J Med. 2013;369(2):134-44

Inman BA, Sebo TJ, Frigola X, et al: PD-L1 (B7-H1) expression by urothelial carcinoma of the bladder and BCG-induced granulomata: associations with localized stage progression. Cancer. 2007;109(8):1499-505

Jarow JP, Lerner SP, Kluetz PG, et al: Clinical trial design for the development of new therapies for nonmuscle-invasive bladder cancer: report of a Food and Drug Administration and American Urological Association public workshop. Urology. 2014; 83(2):262-4

Jung SH, Lee TY, Kim KM, George S (2004). Admissible two-stage designs for phase II cancer clinical trials, Statistics in Medicine 23: 561-569.

Kaehler et al. Update on immunologic therapy with anti-CTLA-4 antibodies in melanoma: identification of clinical and biological response patterns, immune-related adverse events, and their management. <u>Semin Oncol.</u> 2010 Oct;37(5):485-98

Kandalaft LE, Motz GT, Duraiswamy J, et al: Tumor immune surveillance and ovarian cancer: lessons on immune mediated tumor rejection or tolerance. Cancer Metastasis Rev 2011; 30:141-51.

Katsumata N, Yasuda M, Takahashi F, et al: Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet 2009; 374:1331-8.

Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704.

Kim KW, Ramaiya NH, Krajewski KM, et al. Ipilimumab associated hepatitis: imaging and clinicopathologic findings. Invest New Drugs. 2013;31:1071.

Krambeck AE, Dong H, Thompson RH, Kuntz SM, Lohse CM, Leibovich BC, et al: Survivin and B7-H1 are collaborative predictors of survival and represent potential therapeutic targets for patients with renal cell carcinoma. Clin Cancer Res. 2007;13(6):1749-56.

Kryczek I, Wei S, Zhu G, et al: Relationship between B7-H4, regulatory T cells, and patient outcome in human ovarian carcinoma. Cancer Res 2007; 67:8900-5.

Lam JS, Benson MC, O'Donnell MA, et al: Bacillus Calmete-Guérin plus interferon-alpha2B intravesical therapy maintains an extended treatment plan for superficial bladder cancer with minimal toxicity. Urol Oncol. 2003; 21(5):354-60

Lenz. Management and preparedness for infusion and hypersensitivity reactions. <u>Oncologist.</u> 2007;12(5):601-9.

Loos M, Giese NA, Kleeff J, Giese T, Gaida MM, Bergmann F, et al. Clinical significance and regulation of the costimulatory molecule B7-H1 in pancreatic adenocarcinoma. Cancer Lett. 2008;268(1):98-109.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

Mu CY, Huang JA, Chen Y, Chen C, Zhang XG. High expression of PD-L1 in lung cancer may contribute to poor prognosis and tumor cells immune escape through suppressing tumor infiltrating dendritic cells maturation. Med Oncol. 2011 Sep;28(3):682-8.

Nishino M, Giobbie-Hurder A, Gargano M, Suda M, Ramaiya NH and Hodi FS. Developing a common language for tumor response to immunotherapy: immune-related response criteria using unidimensional measurements. Clin Cancer Res. 2013 Jul; 19(14):3936-3943.

Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, et al. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic adenocarcinoma. Clin Cancer Res. 2007 Apr 1;13(7):2151-7.

Park J, Omiya R, Matsumura Y, Sakoda Y, Kuramasu A, Augustine MM, et al. B7-H1/CD80 interaction is required for the induction and maintenance of peripheral T-cell tolerance. Blood. 2010;116(8):1291-8.

Perren TJ, Swart AM, Pfisterer J, et al: A phase 3 trial of bevacizumab in ovarian cancer. The New England journal of medicine 2011; 365:2484-96.

Powles T, Eder JP, Fine GD, et al: MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014;515(7528):558-62.

Raja FA, Chopra N, Ledermann JA. Optimal first-line treatment in ovarian cancer. Ann Oncol 2012 Sep; 23 Suppl 10:x118-27.

Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2015. CA Cancer J Clin 2015 Jan-Feb; 65(1): 5-29.

Simon R (1989). Controlled Clinical Trials 10: 1-10.

Sznol M and Chen L. Antagonist antibodies to PD-1 and B7-H1 (PD-L1) in the treatment of advanced human cancer. 2013; 19(5):1021-1034.

Tarhini A. Immune-mediated adverse events associated with ipilimumab ctla-4 blockade therapy: the underlying mechanisms and clinical management. <u>Scientifica (Cairo)</u>. 2013;2013:857519

TCGA. Integrated genomic analyses of ovarian carcinoma. Nature 2011; 474:609-15.

Thall PF, Simon R. Practical Bayesian guideline for phase IIB clinical trials. Biometrics 1994 Jun;50(2):337-49.

Thall PF, Wooten LH, and Tannir NM. Monitoring Event Times in Early Phase Clinical Trials: Some Practical Issues, Clinical Trials 2005; 2, 467-478 (2005).

Thompson RH, Gillett MD, Chevillem JC, Lohsem CM, Dong H, Webster WS, et al. Costimulatory molecule B7-H1 in primary and metastatic clear cell renal cell carcinoma. Cancer. 2005;104(10):2084-91.

Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, et al. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006;66(7):3381-5.

Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, et al. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54.

US Department of Health and Human Services, National Institutes of Health, National Cancer Institute. Common Terminology Criteria for Adverse Events Version 4.03. http://evs.nci.nih.gov/ftp1/CTCAE/About.html

Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RHM, van der Burg MEL, Lacave AJ, Bendetti Panici P, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GCE, Pecorelli S, Reed NS. Neoadjuvant Chemotherapy or Primary Surgery in Stage IIIc or IV Ovarian Cancer. NEJM 2010; 363; 10: 943-53.

Wang L, Ma Q, Chen X, Guo K, Li J, Zhang M. Clinical significance of B7-H1 and B7-1 expressions in pancreatic carcinoma. World J Surg. 2010;34(5):1059-65.

Weber et al. Management of immune-related adverse events and kinetics of response with ipilimumab. <u>J Clin Oncol.</u> 2012 Jul 20;30(21):2691-7

Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbé, et al. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009;15:7412-20.

Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008;8(6):467-77.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

# Dosing Modification and Toxicity Management Guidelines for Immune-Mediated, Infusion-Related, and

# Non-Immune–Mediated Reactions (MEDI4736 Monotherapy or Combination Therapy With Tremelimumab or Tremelimumab Monotherapy) 1 November 2017 Version

## **General Considerations**

#### **Dose Modifications**

Drug administration modifications of study drug/study regimen will be made to manage potential immune-related AEs based on severity of treatment-emergent toxicities graded per NCI CTCAE v4.03.

In addition to the criteria for permanent discontinuation of study drug/study regimen based on CTC grade/severity (table below), permanently discontinue study drug/study regimen for the following conditions:

- Inability to reduce corticosteroid to a dose of ≤10 mg of prednisone per day (or equivalent) within 12 weeks after last dose of study drug/study regimen
- Recurrence of a previously experienced Grade 3 treatment-related AE following resumption of dosing

Grade 1 No dose modification

Grade 2 Hold study drug/study regimen dose until Grade 2 resolution to Grade  $\leq 1$ .

If toxicity worsens, then treat as Grade 3 or Grade 4.

Study drug/study regimen can be resumed once event stabilizes to Grade ≤1 after completion of steroid taper.

Patients with endocrinopathies who may require prolonged or continued steroid replacement can be retreated with study drug/study regimen on the following

## conditions:

- 1. The event stabilizes and is controlled.
- The patient is clinically stable as per Investigator or treating physician's clinical judgement.
- 3. Doses of prednisone are at ≤10 mg/day or equivalent.

Grade 3 Depending on the individual toxicity, study drug/study regimen may be permanently

#### **Toxicity Management**

It is recommended that management of immune-mediated adverse events (imAEs) follows the guidelines presented in this table:

- It is possible that events with an inflammatory or immune mediated mechanism could occur in nearly all organs, some of them not noted specifically in these guidelines.
- Whether specific immune-mediated events (and/or laboratory indicators of such events) are noted in these guidelines or not, patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression, concomitant medications, and infections) to a possible immune-mediated event. In the absence of a clear alternative etiology, all such events should be managed as if they were immune related. General recommendations follow.
- Symptomatic and topical therapy should be considered for low-grade (Grade 1 or 2, unless otherwise specified) events.
- For persistent (>3 to 5 days) low-grade (Grade 2) or severe (Grade ≥3) events, promptly start prednisone 1 to 2 mg/kg/day PO or IV equivalent.
- Some events with high likelihood for morbidity and/or mortality e.g., myo-carditis, or other similar events even if they are not currently noted in the guidelines should progress rapidly to high dose IV corticosteroids (methylprednisolone at 2 to 4 mg/kg/day) even if the event is Grade 2, and if clinical suspicion is high and/or there has been clinical confirmation. Consider, as necessary, discussing with the study physician, and promptly pursue specialist consultation.
- If symptoms recur or worsen during corticosteroid tapering (28 days of taper), increase the corticosteroid dose (prednisone dose [e.g., up to 2 to 4 mg/kg/day PO or IV equivalent]) until stabilization or improvement of symptoms, then resume corticosteroid tapering at a slower rate (>28 days of taper).
- More potent immunosuppressives such as TNF inhibitors (e.g., infliximab) (also refer to the individual sections of the imAEs for specific type of immunosuppressive) should be considered for events not responding to systemic steroids.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

# Dosing Modification and Toxicity Management Guidelines for Immune-Mediated, Infusion-Related, and

# Non-Immune–Mediated Reactions (MEDI4736 Monotherapy or Combination Therapy With Tremelimumab or Tremelimumab Monotherapy) 1 November 2017 Version

## **General Considerations**

#### **Dose Modifications Toxicity Management** Progression to use of more potent discontinued. Please refer to guidelines below. immunosuppressives should proceed more Grade 4 Permanently discontinue study drug/study rapidly in events with high likelihood for morbidity and/or mortality - e.g., myocarditis, or regimen. other similar events even if they are not currently Note: For Grade ≥3 asymptomatic amylase or lipase levels, noted in the guidelines – when these events are hold study drug/study regimen, and if complete work up not responding to systemic steroids. With long-term steroid and other shows no evidence of pancreatitis, study drug/study regimen immunosuppressive use, consider need for may be continued or resumed. Pneumocystis jirovecii pneumonia (PJP, formerly Note: Study drug/study regimen should be permanently known as Pneumocystis carinii pneumonia) prophylaxis, gastrointestinal protection, and discontinued in Grade 3 events with high likelihood for glucose monitoring. morbidity and/or mortality - e.g., myocarditis, or other similar Discontinuation of study drug/study regimen is events even if they are not currently noted in the guidelines. not mandated for Grade 3/Grade 4 inflammatory reactions attributed to local tumor response Similarly, consider whether study drug/study regimen should (e.g., inflammatory reaction at sites of metastatic be permanently discontinued in Grade 2 events with high disease and lymph nodes). Continuation of study likelihood for morbidity and/or mortality - e.g., myocarditis, drug/study regimen in this situation should be based upon a benefit-risk analysis for that patient. or other similar events even if they are not currently noted in the guidelines – when they do not rapidly improve to Grade <1 upon treatment with systemic steroids and following full taper Note: There are some exceptions to permanent discontinuation of study drug for Grade 4 events (i.e., hyperthyroidism, hypothyroidism, Type 1 diabetes mellitus).

AE Adverse event; CTC Common Toxicity Criteria; CTCAE Common Terminology Criteria for Adverse Events; imAE immune-mediated adverse event; IV intravenous; NCI National Cancer Institute; PO By mouth.

| Pediatric Considerations | |
|---|---|
| <b>Dose Modifications</b> | Toxicity Management |
| The criteria for permanent discontinuation of study drug/study regimen based on CTC grade/severity is the | <ul> <li>All recommendations for specialist consultation<br/>should occur with a pediatric specialist in the<br/>specialty recommended.</li> </ul> |
| same for pediatric patients as it is for adult patients, as well as to permanently discontinue study drug/study regimen if unable to reduce corticosteroid ≤ a dose | <ul> <li>The recommendations for dosing of steroids (i.e.,<br/>mg/kg/day) and for IV IG and plasmapheresis that are<br/>provided for adult patients should also be used for<br/>pediatric patients.</li> </ul> |

Clinical Study Protocol
Drug Substance Durvalumab (Medi4736)
Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

| Pediatric Considerations | |
|---|---|
| Dose Modifications | Toxicity Management |
| equivalent to that required for corticosteroid replacement therapy within 12 weeks after last dose of study drug/study regimen | <ul> <li>The infliximab 5 mg/kg IV dose recommended for adults is the same as recommended for pediatric patients ≥ 6 years old. For dosing in children younger than 6 years old, consult with a pediatric specialist.</li> </ul> |
| | <ul> <li>For pediatric dosing of mycophenolate mofetil,<br/>consult with a pediatric specialist.</li> </ul> |
| | <ul> <li>With long-term steroid and other immunosuppressive<br/>use, consider need for PJP prophylaxis,<br/>gastrointestinal protection, and glucose monitoring.</li> </ul> |

Edition Number 1.9.4

Date 10/08/2018

# **Specific Immune-Mediated Reactions**

| Adverse Events | Severity Grade<br>of the Event<br>(NCI CTCAE<br>version 4.03) | Dose Modifications | Toxicity Management |
|---|---|---|---|
| Pneumonitis/Interstitial Lung Disease (ILD) | Any Grade | General Guidance | For Any Grade: - Monitor patients for signs and symptoms of pneumonitis or ILD (new onset or worsening shortness of breath or cough). Patients should be evaluated with imaging and pulmonary function tests, including other diagnostic procedures as described below. - Initial work-up may include clinical evaluation, monitoring of oxygenation via pulse oximetry (resting and exertion), laboratory work-up, and high- resolution CT scan. |
| | Grade 1 (asymptomatic, clinical or diagnostic observations only; intervention not indicated) | No dose modifications<br>required. However,<br>consider holding study<br>drug/study regimen dose<br>as clinically appropriate<br>and during diagnostic<br>work-up for other<br>etiologies. | For Grade 1 (radiographic changes only): - Monitor and closely follow up in 2 to 4 days for clinical symptoms, pulse oximetry (resting and exertion), and laboratory work-up and then as clinically indicated. - Consider Pulmonary and Infectious disease consult. |
| | Grade 2 (symptomatic; medical intervention indicated; limiting instrumental ADL) | Hold study drug/study regimen dose until Grade 2 resolution to Grade ≤1. If toxicity worsens, then treat as Grade 3 or Grade 4. If toxicity improves to Grade ≤1, then the decision to reinitiate study drug/study regimen will be based upon treating physician's clinical judgment and after completion of steroid taper. | For Grade 2 (mild to moderate new symptoms): - Monitor symptoms daily and consider hospitalization. - Promptly start systemic steroids (e.g., prednisone 1 to 2 mg/kg/day PO or IV equivalent). - Reimage as clinically indicated. - If no improvement within 3 to 5 days, additional workup should be considered and prompt treatment with IV methylprednisolone 2 to 4 mg/kg/day started - If still no improvement within 3 to 5 days despite IV methylprednisolone at 2 to 4 mg/kg/day, promptly start immunosuppressive therapy such as TNF inhibitors (e.g., infliximab at 5 mg/kg every 2 weeks). Caution: It is important to rule out sepsis and |

Edition Number 1.9.4

| e 10/06/2016 | | | |
|---|---|---|---|
| | | | refer to infliximab label for general guidance before using infliximab. |
| | | | <ul> <li>Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, or anti-PJP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation])<sup>a</sup></li> </ul> |
| | | | <ul> <li>Consider pulmonary and infectious disease consult.</li> </ul> |
| | | | <ul> <li>Consider, as necessary, discussing with study physician.</li> </ul> |
| | Grade 3 or 4 | Permanently discontinue | For Grade 3 or 4 (severe or new symptoms |
| | (Grade 3: severe | study drug/study regimen. | new/worsening hypoxia, life-threatening): |
| | symptoms;<br>limiting self-care | | <ul> <li>Promptly initiate empiric IV<br/>methylprednisolone 1 to 4 mg/kg/da<br/>or equivalent.</li> </ul> |
| | ADL; oxygen indicated) | | <ul> <li>Obtain Pulmonary and Infectious<br/>disease consult; consider, as<br/>necessary, discussing with study<br/>physician.</li> </ul> |
| | (Grade 4: life- | | <ul> <li>Hospitalize the patient.</li> </ul> |
| | threatening | | <ul> <li>Supportive care (e.g., oxygen).</li> </ul> |
| | respiratory<br>compromise;<br>urgent<br>intervention<br>indicated [e.g.,<br>tracheostomy or<br>intubation]) | | <ul> <li>If no improvement within 3 to 5 days, additional workup should be considered and prompt treatment with additional immunosuppressive therapy such as TNF inhibitors (e.g., infliximab at 5 mg/kg every 2 weeks' dose) started. Caution: rule out sepsis and refer to infliximab label for general guidance before using infliximab.</li> </ul> |
| | | | <ul> <li>Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and, in particular, anti-PJP treatment (refer to current NCCN guidelines for treatment of cancer-related infection [Category 2B recommendation]).<sup>a</sup></li> </ul> |
| Diarrhea/Colitis | Any Grade | General Guidance | For Any Grade: |
| | | | <ul> <li>Monitor for symptoms that may be related to diarrhea/enterocolitis <ul> <li>(abdominal pain, cramping, or changes in bowel habits such as increased frequency over baseline o blood in stool) or related to bowel perforation (such as sepsis, peritoneal signs, and ileus).</li> </ul> </li> </ul> |

Edition Number 1.9.4

| | | <ul> <li>Patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression, other medications, or infections), including testing for clostridium difficile toxin, etc.</li> <li>Steroids should be considered in the absence of clear alternative etiology, even for low-grade events, in order to prevent potential progression to higher grade event.</li> <li>Use analgesics carefully; they can mask symptoms of perforation and</li> </ul> |
|---|---|---|
| | | peritonitis. |
| Grade 1 (Diarrhea: stool frequency of <4 over baseline per day) (Colitis: asymptomatic; clinical or diagnostic observations only) | No dose modifications. | For Grade 1: - Monitor closely for worsening symptoms. - Consider symptomatic treatment, including hydration, electrolyte replacement, dietary changes (e.g., American Dietetic Association colitis diet), and loperamide. Use probiotics as per treating physician's clinical judgment. |
| Grade 2 | Hold study drug/study | For Grade 2: |
| (Diarrhea: stool<br>frequency of 4 to<br>6 over baseline<br>per day) (Colitis:<br>abdominal pain;<br>mucus or blood<br>in stool) | regimen until resolution to Grade ≤1 If toxicity worsens, then treat as Grade 3 or Grade 4. If toxicity improves to Grade ≤1, then study drug/study regimen can be resumed after completion of steroid taper. | <ul> <li>Consider symptomatic treatment, including hydration, electrolyte replacement, dietary changes (e.g., American Dietetic Association colitis diet), and loperamide and/or budesonide.</li> <li>Promptly start prednisone 1 to 2 mg/kg/day PO or IV equivalent.</li> <li>If event is not responsive within 3 to 5 days or worsens despite prednisone at 1 to 2 mg/kg/day PO or IV equivalent, GI consult should be obtained for consideration of further workup, such as imaging and/or colonoscopy, to confirm colitis and rule out perforation, and prompt treatment with IV methylprednisolone 2 to 4 mg/kg/day started.</li> <li>If still no improvement within 3 to 5 days despite 2 to 4 mg/kg/IV</li> </ul> |
| | | days despite 2 to 4 mg/kg IV<br>methylprednisolone, promptly start<br>immunosuppressives such as<br>infliximab at 5 mg/kg once every 2 |

Edition Number 1.9.4

Hepatitis (elevated LFTs)

| | | weeks <sup>a</sup> . Caution: it is important to rule out bowel perforation and refer to infliximab label for general guidance before using infliximab. Consider, as necessary, discussing with study physician if no resolution to Grade ≤1 in 3 to 4 days. Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJF treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]). <sup>a</sup> |
|---|---|---|
| Grade 3 or 4 | Grade 3 | For Grade 3 or 4: |
| (Grade 3<br>diarrhea: stool<br>frequency of ≥7<br>over baseline per<br>day; | Permanently discontinue<br>study drug/study regimen<br>for Grade 3 if toxicity<br>does not improve to<br>Grade ≤1 within 14 days; | <ul> <li>Promptly initiate empiric IV methylprednisolone 2 to 4 mg/kg/da or equivalent.</li> <li>Monitor stool frequency and volume and maintain hydration.</li> <li>Urgent GI consult and imaging</li> </ul> |
| Grade 4 diarrhea: life threatening consequences) (Grade 3 colitis: severe abdominal pain, change in bowel habits, medi-cal intervention indi-cated, peritoneal signs; Grade 4 colitis: life-threatening consequences, urgent intervention indicated) | study drug/study regimen can be resumed after completion of steroid taper. Grade 4 Permanently discontinue study drug/study regimen. | and/or colonoscopy as appropriate. If still no improvement within 3 to 5 days of IV methylprednisolone 2 to mg/kg/day or equivalent, promptly start further immunosuppressives (e.g., infliximab at 5 mg/kg once every 2 weeks). Caution: Ensure G consult to rule out bowel perforation and refer to infliximab label for general guidance before using infliximab. Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJI treatment (refer to current NCCN guidelines for treatment of cancer-related infections [Category 2B recommendation]). <sup>a</sup> |
| Any Grade | General Guidance | For Any Grade: - Monitor and evaluate liver function test: AST, ALT, ALP, and TB. - Evaluate for alternative etiologies (e.g., viral hepatitis, disease progression, concomitant |

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

| T 01: 1 1 11 11 | | | | | medications). |
|---|---|---|---|---|---|
| Infliximab should not be | C . 1. 1 | | N 1 | | <u> </u> |
| used for management of immune-related hepatitis. PLEASE SEE shaded area immediately below this section to find | Grade 1 (AST or ALT >ULN and ≤3.0×ULN and/or TB > ULN and ≤1.5×ULN) | • | No dose modifications. If it worsens, then treat as Grade 2 event. | - | For Grade 1: Continue LFT monitoring per protocol. |
| guidance for management of "Hepatitis (elevated LFTS)" in HCC patients | Grade 2 (AST or ALT >3.0×ULN and ≤5.0×ULN and/or TB >1.5×ULN and ≤3.0×ULN) | • | Hold study drug/study regimen dose until Grade 2 resolution to Grade ≤1. If toxicity worsens, then treat as Grade 3 or Grade 4. If toxicity improves to Grade ≤1 or baseline, resume study drug/study regimen after completion of steroid taper. | | For Grade 2: Regular and frequent checking of LFTs (e.g., every 1 to 2 days) until elevations of these are improving or resolved. If no resolution to Grade ≤1 in 1 to 2 days, consider, as necessary, discussing with study physician. If event is persistent (>3 to 5 days) or worsens, promptly start prednisone 1 to 2 mg/kg/day PO or IV equivalent. If still no improvement within 3 to 5 days despite 1 to 2 mg/kg/day of prednisone PO or IV equivalent, consider additional work up and start prompt treatment with IV methylprednisolone 2 to 4 mg/kg/day. If still no improvement within 3 to 5 days despite 2 to 4 mg/kg/day of IV methylprednisolone, promptly start immunosuppressives (i.e., mycophenolate mofetil). Discuss with study physician if mycophenolate mofetil is not available. Infliximab should NOT be used. Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancer- |
| | Grade 3 or 4 | | For Grade 3: | | related infections [Category 2B recommendation]). <sup>a</sup> For Grade 3 or 4: |
| | or ALT >5.0×ULN and ≤20.0×ULN | For elevations in transaminases $\leq 8 \times \text{ULN}$ , or elevations in bilirubin $\leq 5 \times \text{ULN}$ : | ansaminases $\leq 8 \times \text{ULN}$ , or elevations in bilirubin $\leq 5 \times \text{ULN}$ : | _ | Promptly initiate empiric IV methylprednisolone at 1 to 4 mg/kg/day or equivalent. If still no improvement within 3 to 5 days despite 1 to 4 mg/kg/day methylprednisolone IV or equivalent, |
| | and/or | • | Hold study | | 1 |

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

TB >3.0×ULN and  $\leq 10.0 \times ULN$ )

(Grade 4: AST or ALT >20×ULN and/or TB >10×ULN)

- drug/study regimen dose until resolution to Grade ≤1 or baseline
- Resume study drug/study regimen if elevations downgrade to Grade ≤1 or baseline within 14 days and after completion of steroid taper.
- Permanently discontinue study drug/study regimen if the elevations do not downgrade to Grade ≤1 or baseline within 14 days

For elevations in transaminases >8 × ULN or elevations in bilirubin >5 × ULN, discontinue study drug/study regimen.

Permanently discontinue study drug/study regimen for any case meeting Hy's law criteria (AST and/or ALT >3 × ULN + bilirubin >2 × ULN without initial findings of cholestasis (i.e., elevated alkaline P04) and in the absence of any alternative cause.<sup>b</sup>

- promptly start treatment with immunosuppressive therapy (i.e., mycophenolate mofetil). Discuss with study physician if mycophenolate is not available. **Infliximab should NOT be used.**
- Perform hepatology consult, abdominal workup, and imaging as

appropriate.

Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]).<sup>a</sup>

### For Grade 4:

Permanently discontinue study drug/study regimen.

| Hepatitis | Any Grade | General Guidance | For Any Grade: |
|---|---|---|---|
| (elevated LFTs) | | | <ul> <li>Monitor and evaluate liver function<br/>test: AST, ALT, ALP, and TB.</li> </ul> |
| | | | <ul> <li>Evaluate for alternative etiologies <ul> <li>(e.g., viral hepatitis, disease</li> <li>progression, concomitant</li> </ul> </li> </ul> |

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

Infliximab should not be used for management of immune-related hepatitis.

THIS shaded area is guidance *only* for management of "Hepatitis (elevated LFTs)" in HCC patients

See instructions at bottom of shaded area if transaminase rise is not isolated but (at any time) occurs in setting of either increasing bilirubin or signs of DILI/liver decompensation

- medications, worsening of liver cirrhosis [e.g., portal vein thrombosis]).
- For HBV+ patients: evaluate quantitative HBV viral load, quantitative HBsAg, or HBeAg
- For HCV+ patients: evaluate quantitative HCV viral load
- Consider consulting
   hepatologist/Infectious disease
   specialist regarding
   change/implementation in/of
   antiviral medications for any patient
   with an elevated HBV viral load
   >2000 IU/ml
- Consider consulting
   hepatologist/Infectious disease
   specialist regarding
   change/implementation in/of
   antiviral HCV medications if HCV
   viral load increased by ≥2-fold
- For HCV+ with HBcAB+: Evaluate for both HBV and HCV as above

#### Grade 1

(Isolated AST or ALT >ULN and ≤5.0×ULN, whether normal or elevated at baseline)

- No dose modifications.
  - If ALT/AST elevations represents significant worsening based on investigator assessment, then treat as Grade 2 event.

For all grades, see
instructions at bottom of
shaded area if
transaminase rise is not
isolated but (at any time)
occurs in setting of either
increasing bilirubin or
signs of DILI/liver

(Isolated AST or ALT >5.0 $\times$ ULN and  $\leq$ 8.0 $\times$ ULN, if normal at

Grade 2

Hold study drug/study regimen dose until Grade 2 resolution to Grade ≤1 or baseline.

decompensation

### For Grade 2:

- Regular and frequent checking of LFTs (e.g., every 1 to 3 days) until elevations of these are improving or resolved.
- Recommend consult hepatologist;

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

- 10/00/2010

| Date 10/08/2018 | | | |
|---|---|---|---|
| | baseline) | • If toxicity worsens,<br>then treat as Grade 3<br>or Grade 4. | consider abdominal ultrasound, including Doppler assessment of liver perfusion. |
| | (Isolated AST or ALT >2.0×baseline and ≤12.5×ULN, if elevated >ULN at baseline) | If toxicity improves to Grade ≤1 or baseline, resume study drug/study regimen after completion of steroid taper. | <ul> <li>Consider, as necessary, discussing with study physician.</li> <li>If event is persistent (&gt;3 to 5 days) or worsens, and investigator suspects toxicity to be immune-mediated AE, recommend to start prednisone 1 to 2 mg/kg/day PO or IV equivalent.</li> <li>If still no improvement within 3 to 5 days despite 1 to 2 mg/kg/day of prednisone PO or IV equivalent, consider additional workup and treatment with IV methylprednisolone 2 to 4 mg/kg/day.</li> <li>If still no improvement within 3 to 5 days despite 2 to 4 mg/kg/day of IV methylprednisolone, consider additional abdominal workup (including liver biopsy) and imaging (i.e., liver ultrasound), and consider starting immunosuppressives (i.e., mycophenolate mofetil). Discuss with study physician if mycophenolate mofetil is not available. Infliximab should NOT be used.</li> </ul> |
| | Grade 3 (Isolated AST or ALT >8.0×ULN and ≤20.0×ULN, if normal at baseline) (Isolated AST or ALT >12.5×ULN and ≤20.0×ULN, if elevated >ULN at baseline) | <ul> <li>Hold study drug/study regimen dose until resolution to Grade ≤1 or baseline</li> <li>Resume study drug/study regimen if elevations downgrade to Grade ≤1 or baseline within 14 days and after completion of steroid taper.</li> <li>Permanently discontinue study drug/study regimen if the elevations do not downgrade to Grade ≤1 or baseline within 14 days</li> <li>Permanently discontinue study drug/study regimen if the elevations do not downgrade to Grade ≤1 or baseline within 14 days</li> <li>Permanently discontinue study drug/study regimen for any case meeting Hy's</li> </ul> | For Grade 3: Regular and frequent checking of LFTs (e.g., every 1-2 days) until elevations of these are improving or resolved. Consult hepatologist (unless investigator is hepatologist); obtain abdominal ultrasound, including Doppler assessment of liver perfusion; and consider liver biopsy. Consider, as necessary, discussing with study physician. If investigator suspects toxicity to be immune-mediated, promptly initiate empiric IV methylprednisolone at 1 to 4 mg/kg/day or equivalent. If no improvement within 3 to 5 days despite 1 to 4 mg/kg/day methylprednisolone IV or equivalent, obtain liver biopsy (if it has not been done already) and promptly start treatment with immunosuppressive therapy (mycophenolate mofetil). Discuss with study physician if |

Clinical Study Protocol Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

| | law criteria, in the<br>absence of any alternative<br>cause. <sup>b</sup> | mycophenolate is not available. Infliximab should NOT be used. Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PCP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]). <sup>a</sup> |
|---|---|---|
| Grade 4 | Permanently discontinue | For Grade 4: |
| (Isolated AST or | study drug/study regimen. | Same as above |
| ALT >20×ULN, | | (except would recommend obtaining liver |
| whether normal | | biopsy early) |
| or elevated at | | |
| baseline) | | |

If transaminase rise is not isolated but (at any time) occurs in setting of either increasing total/direct bilirubin ( $\geq$ 1.5×ULN, if normal at baseline; or 2×baseline, if >ULN at baseline) or signs of DILI/liver decompensation (e.g., fever, elevated INR):

- Manage dosing for Grade 1 transaminase rise as instructed for Grade 2 transaminase rise
- Manage dosing for Grade 2 transaminase rise as instructed for Grade 3 transaminase rise
- Grade 3-4: Permanently discontinue study drug/study regimen

| Nephritis or renal | Any Grade | General Guidance | For Any Grade: |
|---|---|---|---|
| dysfunction | | | <ul> <li>Consult with nephrologist.</li> </ul> |
| (elevated serum creatinine) | | | <ul> <li>Monitor for signs and symptoms that<br/>may be related to changes in renal<br/>function (e.g., routine urinalysis,<br/>elevated serum BUN and creatinine,<br/>decreased creatinine clearance,<br/>electrolyte imbalance, decrease in<br/>urine output, or proteinuria).</li> </ul> |
| | | | <ul> <li>Patients should be thoroughly<br/>evaluated to rule out any alternative<br/>etiology (e.g., disease progression or<br/>infections).</li> </ul> |
| | | | <ul> <li>Steroids should be considered in the<br/>absence of clear alternative etiology<br/>even for low-grade events (Grade 2),<br/>in order to prevent potential<br/>progression to higher grade event.</li> </ul> |
| | Grade 1 | No dose modifications. | For Grade 1: |

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

| | | M 5 2 11 1 |
|---|---|---|
| (Serum | | <ul> <li>Monitor serum creatinine weekly and any accompanying symptoms.</li> </ul> |
| creatinine > 1 to<br>1.5 × baseline; ><br>ULN to 1.5 ×<br>ULN) | | <ul> <li>If creatinine returns to<br/>baseline, resume its regular<br/>monitoring per study<br/>protocol.</li> </ul> |
| OLIV | | • If creatinine worsens, depending on the severity, treat as Grade 2, 3, or 4. |
| | | <ul> <li>Consider symptomatic treatment,<br/>including hydration, electrolyte<br/>replacement, and diuretics.</li> </ul> |
| Grade 2 | Hold study drug/study | For Grade 2: |
| regimen until resolution to Grade ≤1 or baseline. to 3.0 × baseline; >1.5 to 3.0 × ULN) • If toxicity worsens, then treat as Grade 3 or 4. • If toxicity improves to Grade ≤1 or baseline, then resume study drug/study regimen after completion of steroid taper. | <ul> <li>Consider symptomatic treatment,<br/>including hydration, electrolyte<br/>replacement, and diuretics.</li> </ul> | |
| | <ul> <li>Carefully monitor serum creatinine<br/>every 2 to 3 days and as clinically<br/>warranted.</li> </ul> | |
| | <ul> <li>Consult nephrologist and consider<br/>renal biopsy if clinically indicated.</li> </ul> | |
| | study drug/study<br>regimen after | <ul> <li>If event is persistent (&gt;3 to 5 days) or<br/>worsens, promptly start prednisone 1<br/>to 2 mg/kg/day PO or IV equivalent.</li> </ul> |
| | <ul> <li>If event is not responsive within 3 to<br/>5 days or worsens despite prednisone<br/>at 1 to 2 mg/kg/day PO or IV<br/>equivalent, additional workup should<br/>be considered and prompt treatment<br/>with IV methylprednisolone at 2 to<br/>4 mg/kg/day started.</li> </ul> | |
| | | <ul> <li>Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]).<sup>a</sup></li> </ul> |
| | | <ul> <li>When event returns to baseline,<br/>resume study drug/study regimen and<br/>routine serum creatinine monitoring<br/>per study protocol.</li> </ul> |
| Grade 3 or 4 | Permanently discontinue | For Grade 3 or 4: |
| (Grade 3: serum | study drug/study regimen. | <ul> <li>Carefully monitor serum creatinine<br/>on daily basis.</li> </ul> |
| creatinine >3.0 × baseline; | | <ul> <li>Consult nephrologist and consider<br/>renal biopsy if clinically indicated.</li> </ul> |
| $>3.0$ to $6.0 \times ULN$ ; | | <ul> <li>Promptly start prednisone 1 to 2<br/>mg/kg/day PO or IV equivalent.</li> </ul> |
| | | <ul> <li>If event is not responsive within 3 to</li> <li>5 days or worsens despite prednisone</li> </ul> |

Edition Number 1.9.4

| | Grade 4: serum<br>creatinine >6.0 ×<br>ULN) | | at 1 to 2 mg/kg/day PO or IV equivalent, additional workup should be considered and prompt treatment with IV methylprednisolone 2 to 4 mg/kg/day started. - Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]). <sup>a</sup> |
|---|---|---|---|
| Rash (excluding bullous skin formations) | Any Grade (refer to NCI CTCAE v 4.03 for definition of severity/grade depending on type of skin rash) | General Guidance | For Any Grade: - Monitor for signs and symptoms of dermatitis (rash and pruritus). - IF THERE IS ANY BULLOUS FORMATION, THE STUDY PHYSICIAN SHOULD BE CONTACTED AND STUDY DRUG DISCONTINUED. |
| | Grade 1 | No dose modifications. | For Grade 1: - Consider symptomatic treatment, including oral antipruritics (e.g., diphenhydramine or hydroxyzine) and topical therapy (e.g., urea cream). |
| | Grade 2 | For persistent (>1 to 2 weeks) Grade 2 events, hold scheduled study drug/study regimen until resolution to Grade ≤1 or baseline. If toxicity worsens, then treat as Grade 3. If toxicity improves to Grade ≤1 or baseline, then resume drug/study regimen after completion of steroid taper. | For Grade 2: Obtain dermatology consult. Consider symptomatic treatment, including oral antipruritics (e.g., diphenhydramine or hydroxyzine) and topical therapy (e.g., urea cream). Consider moderate-strength topical steroid. If no improvement of rash/skin lesions occurs within 3 to 5 days or is worsening despite symptomatic treatment and/or use of moderate strength topical steroid, consider, as necessary, discussing with study physician and promptly start systemic steroids such as prednisone 1 to 2 mg/kg/day PO or IV equivalent. Consider skin biopsy if the event is persistent for >1 to 2 weeks or |

Edition Number 1.9.4

Date 10/08/2018

| recurs. |
|---------|
|---------|

Consider, as necessary, discussing

with study physician.

#### Grade 3 or 4 For Grade 3: For Grade 3 or 4: Consult dermatology. Hold study drug/study Promptly initiate empiric IV regimen until resolution methylprednisolone 1 to 4 mg/kg/day to Grade ≤1 or baseline. or equivalent. Consider hospitalization. If temporarily holding the Monitor extent of rash [Rule of study drug/study regimen Nines]. does not provide Consider skin biopsy (preferably improvement of the Grade more than 1) as clinically feasible. 3 skin rash to Grade ≤1 or Once the patient is improving, gradually taper steroids over ≥28 baseline within 30 days, days and consider prophylactic then permanently antibiotics, antifungals, and anti-PJP discontinue study treatment (refer to current NCCN guidelines for treatment of cancerdrug/study regimen. related infections [Category 2B recommendation]).a

| Endocrinopathy | Any Grade | General Guidance | For Any Grade: |
|---|---|---|---|
| (e.g., hyperthyroidism, | (depending on | | <ul> <li>Consider consulting an endocrinologist for endocrine events.</li> </ul> |
| hypothyroidism, Type 1 diabetes mellitus, | the type of endocrinopathy, | | <ul> <li>Consider, as necessary, discussing with study physician.</li> </ul> |
| hypophysitis, hypopituitarism, and adrenal insufficiency; exocrine event of amylase/lipase increased also included in this | refer to NCI CTCAE v4.03 for defining the CTC grade/severity) | | <ul> <li>Monitor patients for signs and<br/>symptoms of endocrinopathies. Non-<br/>specific symptoms include headache,<br/>fatigue, behavior changes, changed<br/>mental status, vertigo, abdominal<br/>pain, unusual bowel habits,<br/>polydipsia, polyuria, hypotension,<br/>and weakness.</li> </ul> |
| section) | | | Patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression including brain metastases, or infections). |
| | | | <ul> <li>Depending on the suspected<br/>endocrinopathy, monitor and<br/>evaluate thyroid function tests: TSH,<br/>free T3 and free T4 and other<br/>relevant endocrine and related labs<br/>(e.g., blood glucose and ketone<br/>levels, HgA1c).</li> </ul> |

For Grade 4:

Permanently discontinue study drug/study regimen.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- For modest asymptomatic elevations in serum amylase and lipase, corticosteroid treatment is not indicated as long as there are no other signs or symptoms of pancreatic inflammation.
- If a patient experiences an AE that is thought to be possibly of autoimmune nature (e.g., thyroiditis, pancreatitis, hypophysitis, or diabetes insipidus), the investigator should send a blood sample for appropriate autoimmune antibody testing.

#### Grade 1

No dose modifications.

# For Grade 1 (including those with asymptomatic TSH elevation):

- Monitor patient with appropriate endocrine function tests.
- For suspected hypophysitis/hypopituitarism, consider consultation of an endocrinologist to guide assessment of early-morning ACTH, cortisol, TSH and free T4; also consider gonadotropins, sex hormones, and prolactin levels, as well as cosyntropin stimulation test (though it may not be useful in diagnosing early secondary adrenal insufficiency).
- If TSH < 0.5 × LLN, or TSH >2 × ULN, or consistently out of range in 2 subsequent measurements, include free T4 at subsequent cycles as clinically indicated and consider consultation of an endocrinologist.

#### Grade 2

For Grade 2
endocrinopathy other than
hypothyroidism and Type
1 diabetes mellitus, hold
study drug/study regimen
dose until patient is
clinically stable.

• If toxicity worsens, then treat as Grade 3 or Grade 4.

Study drug/study regimen can be resumed once event stabilizes and after

# For Grade 2 (including those with symptomatic endocrinopathy):

- Consult endocrinologist to guide evaluation of endocrine function and, as indicated by suspected endocrinopathy and as clinically indicated, consider pituitary scan.
- For all patients with abnormal endocrine work up, except those with isolated hypothyroidism or Type 1 DM, and as guided by an endocrinologist, consider short-term corticosteroids (e.g., 1 to 2 mg/kg/day methylprednisolone or IV equivalent) and prompt initiation of treatment with relevant hormone

Edition Number 1.9.4

Date 10/08/2018

completion of steroid taper.

Patients with
endocrinopathies who
may require prolonged or
continued steroid
replacement (e.g., adrenal
insufficiency) can be
retreated with study
drug/study regimen on the
following conditions:

- 1. The event stabilizes and is controlled.
- 2. The patient is clinically stable as per investigator or treating physician's clinical judgement.
- Doses of prednisone are ≤10 mg/day or equivalent.

- replacement (e.g., hydrocortisone, sex hormones).
- Isolated hypothyroidism may be treated with replacement therapy, without study drug/study regimen interruption, and without corticosteroids.
- Isolated Type 1 diabetes mellitus (DM) may be treated with appropriate diabetic therapy, without study drug/study regimen interruption, and without corticosteroids.
- Once patients on steroids are improving, gradually taper immunosuppressive steroids (as appropriate and with guidance of endocrinologist) over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancer-related infections [Category 2B recommendation]).<sup>a</sup>
- For patients with normal endocrine workup (laboratory assessment or MRI scans), repeat laboratory assessments/MRI as clinically indicated.

#### Grade 3 or 4

For Grade 3 or 4 endocrinopathy other than hypothyroidism and Type 1 diabetes mellitus, hold study drug/study regimen dose until endocrinopathy symptom(s) are controlled.

Study drug/study regimen can be resumed once event stabilizes and after completion of steroid

taper.

Patients with
endocrinopathies who
may require prolonged or
continued steroid
replacement (e.g., adrenal
insufficiency) can be

#### For Grade 3 or 4:

- Consult endocrinologist to guide evaluation of endocrine function and, as indicated by suspected endocrinopathy and as clinically indicated, consider pituitary scan. Hospitalization recommended.
- For all patients with abnormal endocrine work up, except those with isolated hypothyroidism or Type 1 DM, and as guided by an endocrinologist, promptly initiate empiric IV methylprednisolone 1 to 2 mg/kg/day or equivalent, as well as relevant hormone replacement (e.g., hydrocortisone, sex hormones).
- For adrenal crisis, severe dehydration, hypotension, or shock, immediately initiate IV corticosteroids with mineralocorticoid activity.
- Isolated hypothyroidism may be treated with replacement therapy, without study drug/study regimen interruption, and without

Edition Number 1.9.4

| | | retreated with study | | corticosteroids. |
|---|---|---|---|---|
| | | drug/study regimen on the | _ | Isolated Type 1 diabetes mellitus may be treated with appropriate |
| | | following conditions: | | diabetic therapy, without study |
| | | 1. The event stabilizes | | drug/study regimen interruption, and |
| | | and is controlled. | | without corticosteroids. |
| | | <ol> <li>The patient is clinically stable as per investigator or treating physician's clinical judgement.</li> <li>Doses of prednisone are ≤10 mg/day or equivalent.</li> </ol> | - | Once patients on steroids are improving, gradually taper immunosuppressive steroids (as appropriate and with guidance of endocrinologist) over ≥28 days and consider prophylactic antibiotics, antifungals, and anti-PJP treatment (refer to current NCCN guidelines for treatment of cancer-related infections [Category 2B recommendation]). <sup>a</sup> |
| Neurotoxicity | Any Grade | General Guidance | | For Any Grade: |
| (to include but not be | (depending on | | _ | Patients should be evaluated to rule |
| limited to limbic | the type of | | | out any alternative etiology (e.g., |
| | | | | disease progression, infections, metabolic syndromes, or |
| encephalitis and | neurotoxicity,<br>refer to NCI | | | medications). |
| autonomic neuropathy, | CTCAE v4.03 | | _ | Monitor patient for general |
| excluding Myasthenia | | | | symptoms (headache, nausea, |
| Gravis and Guillain- | for defining the | | | vertigo, behavior change, or weakness). |
| Barre) | CTC | | _ | Consider appropriate diagnostic |
| | grade/severity) | | | testing (e.g., electromyogram and nerve conduction investigations). |
| | | | _ | Perform symptomatic treatment with neurological consult as appropriate. |
| | | | | _ |
| | Grade 1 | No dose modifications. | | For Grade 1: |
| | | | _ | See "Any Grade" recommendations above. |
| | Grade 2 | For acute motor | | For Grade 2: |
| | | neuropathies or<br>neurotoxicity, hold study | _ | Consider, as necessary, discussing with the study physician. |
| | | drug/study regimen dose | _ | Obtain neurology consult. |
| | | until resolution to Grade | - | Sensory neuropathy/neuropathic pain |
| | | ≤1. | | may be managed by appropriate medications (e.g., gabapentin or |
| | | | | duloxetine). |
| | | For sensory | _ | Promptly start systemic steroids |
| | | neuropathy/neuropathic | | prednisone 1 to 2 mg/kg/day PO or |
| | | pain, consider holding | | IV equivalent. |
| | | study drug/study regimen<br>dose until resolution to | _ | If no improvement within 3 to 5 days despite 1 to 2 mg/kg/day prednisone |
| | | | | PO or IV equivalent, consider |

Clinical Study Protocol Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

| Date 10/08/2018 | | | |
|---|---|---|---|
| _ | | Grade ≤1. | additional workup and promptly treat with additional immunosuppressive |
| | | If toxicity worsens, | therapy (e.g., IV IG). |
| | | then treat as Grade 3 | |
| | | or 4. | |
| | | Study drug/study regimen | |
| | | can be resumed once | |
| | | event improves to Grade ≤1 and after completion | |
| | | of steroid taper. | |
| - | Grade 3 or 4 | For Grade 3: | For Grade 3 or 4: |
| | | Hold study drug/study | <ul> <li>Consider, as necessary, discussing with study physician.</li> </ul> |
| | | regimen dose until<br>resolution to Grade ≤1. | <ul> <li>Obtain neurology consult.</li> </ul> |
| | | Permanently discontinue | - Consider hospitalization. |
| | | study drug/study regimen | <ul> <li>Promptly initiate empiric IV<br/>methylprednisolone 1 to 2 mg/kg/day<br/>or equivalent.</li> </ul> |
| | | if Grade 3 imAE does not resolve to Grade ≤1 | - If no improvement within 3 to 5 days |
| | | within 30 days. | despite IV corticosteroids, consider<br>additional workup and promptly treat<br>with additional immunosuppressants<br>(e.g., IV IG). |
| | | For Grade 4: | <ul><li>Once stable, gradually taper steroids</li></ul> |
| | | Permanently discontinue | over ≥28 days. |
| | | study drug/study regimen. | |
| Peripheral neuromotor | Any Grade | General Guidance | For Any Grade: |
| syndromes (such as Guillain-Barre and myasthenia gravis) | | | <ul> <li>The prompt diagnosis of immune-mediated peripheral neuromotor syndromes is important, since certain patients may unpredictably experience acute decompensations that can result in substantial morbidity or in the worst case, death. Special care should be taken for certain sentinel symptoms that may predict a more severe outcome, such as prominent dysphagia, rapidly progressive weakness, and signs of respiratory insufficiency or autonomic instability.</li> <li>Patients should be evaluated to rule out any alternative etiology (e.g., disease progression, infections, metabolic syndromes or medications). It should be noted that the diagnosis of immune-mediated peripheral neuromotor syndromes can be particularly challenging in patients with underlying cancer, due</li> </ul> |

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- to the multiple potential confounding effects of cancer (and its treatments) throughout the neuraxis. Given the importance of prompt and accurate diagnosis, it is essential to have a low threshold to obtain a neurological consult.
- Neurophysiologic diagnostic testing (e.g., electromyogram and nerve conduction investigations, and "repetitive stimulation" if myasthenia is suspected) are routinely indicated upon suspicion of such conditions and may be best facilitated by means of a neurology consultation.
- It is important to consider that the use of steroids as the primary treatment of Guillain-Barre is not typically considered effective.
   Patients requiring treatment should be started with IV IG and followed by plasmapheresis if not responsive to IV IG.

### Grade 1

No dose modifications.

### For Grade 1:

- Consider, as necessary, discussing with the study physician.
- Care should be taken to monitor patients for sentinel symptoms of a potential decompensation as described above.
- Obtain a neurology consult.

#### Grade 2

Hold study drug/study regimen dose until resolution to Grade <1.

Permanently discontinue study drug/study regimen if it does not resolve to Grade ≤1 within 30 days or if there are signs of respiratory insufficiency or autonomic instability.

#### For Grade 2:

- Consider, as necessary, discussing with the study physician.
- Care should be taken to monitor patients for sentinel symptoms of a potential decompensation as described above.
- Obtain a neurology consult
- Sensory neuropathy/neuropathic pain may be managed by appropriate medications (e.g., gabapentin or duloxetine).

#### MYASTHENIA GRAVIS:

 Steroids may be successfully used to treat myasthenia gravis. It is important to consider that steroid therapy (especially with high doses) may result

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

- in transient worsening of myasthenia and should typically be administered in a monitored setting under supervision of a consulting neurologist.
- Patients unable to tolerate steroids may be candidates for treatment with plasmapheresis or IV IG. Such decisions are best made in consultation with a neurologist, taking into account the unique needs of each patient.
- If myasthenia gravis-like neurotoxicity is present, consider starting AChE inhibitor therapy in addition to steroids. Such therapy, if successful, can also serve to reinforce the diagnosis.

#### GUILLAIN-BARRE:

- It is important to consider here that the use of steroids as the primary treatment of Guillain-Barre is not typically considered effective.
- Patients requiring treatment should be started with IV IG and followed by plasmapheresis if not responsive to IV IG.

#### Grade 3 or 4

#### For Grade 3:

Hold study drug/study regimen dose until resolution to Grade ≤1.

Permanently discontinue study drug/study regimen if Grade 3 imAE does not resolve to Grade ≤1 within 30 days or if there are signs of respiratory insufficiency or autonomic instability.

# For Grade 3 or 4 (severe or life-threatening events):

- Consider, as necessary, discussing with study physician.
- Recommend hospitalization.
- Monitor symptoms and obtain neurological consult.

#### MYASTHENIA GRAVIS:

 Steroids may be successfully used to treat myasthenia gravis. They should typically be administered in a monitored setting under supervision of a consulting neurologist.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

#### For Grade 4:

Permanently discontinue study drug/study regimen.

- Patients unable to tolerate steroids may be candidates for treatment with plasmapheresis or IV IG.
- If myasthenia gravis-like neurotoxicity present, consider starting AChE inhibitor therapy in addition to steroids. Such therapy, if successful, can also serve to reinforce the diagnosis.

#### GUILLAIN-BARRE:

- It is important to consider here that the use of steroids as the primary treatment of Guillain-Barre is not typically considered effective.
- Patients requiring treatment should be started with IV IG and followed by plasmapheresis if not responsive to IV IG.

Myocarditis

Any Grade

## **General Guidance**

Discontinue drug permanently if biopsyproven immune-mediated myocarditis.

### For Any Grade:

- The prompt diagnosis of immunemediated myocarditis is important, particularly in patients with baseline cardiopulmonary disease and reduced cardiac function.
- Consider, as necessary, discussing with the study physician.
- Monitor patients for signs and symptoms of myocarditis (new onset or worsening chest pain, arrhythmia, shortness of breath, peripheral edema). As some symptoms can overlap with lung toxicities, simultaneously evaluate for and rule out pulmonary toxicity as well as other causes (e.g., pulmonary embolism, congestive heart failure, malignant pericardial effusion). A Cardiology consultation should be obtained early, with prompt assessment of whether and when to complete a cardiac biopsy, including any other diagnostic procedures.
- Initial work-up should include clinical evaluation, BNP, cardiac enzymes, ECG, echocardiogram (ECHO), monitoring of oxygenation via pulse oximetry (resting and

Edition Number 1.9.4

| | | exertion), and additional laboratory work-up as indicated. Spiral CT or cardiac MRI can complement ECHO to assess wall motion abnormalities when needed. Patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression, other medications, or infections) |
|---|---|---|
| Grade 1 (asymptomatic with laboratory (e.g., BNP) or cardiac imaging abnormalities) | No dose modifications required unless clinical suspicion is high, in which case hold study drug/study regimen dose during diagnostic work-up for other etiologies. If study drug/study regimen is held, resume after complete resolution to Grade 0. | For Grade 1 (no definitive findings): - Monitor and closely follow up in 2 to 4 days for clinical symptoms, BNP, cardiac enzymes, ECG, ECHO, pulse oximetry (resting and exertion), and laboratory work-up as clinically indicated. - Consider using steroids if clinical suspicion is high. |
| Grade 2, 3 or 4 (Grade 2: Symptoms with mild to moderate activity or exertion) (Grade 3: Severe with symptoms at rest or with minimal activity or exertion; intervention indicated) (Grade 4: Lifethreatening consequences; urgent intervention | - If Grade 2 Hold study drug/study regimen dose until resolution to Grade 0. If toxicity rapidly improves to Grade 0, then the decision to reinitiate study drug/study regimen will be based upon treating physician's clinical judgment and after completion of steroid taper. If toxicity does not rapidly improve, permanently. discontinue study drug/study regimen. If Grade 3-4, permanently | For Grade 2-4: Monitor symptoms daily, hospitalize. Promptly start IV methylprednisolone 2 to 4 mg/kg/day or equivalent after Cardiology consultation has determined whether and when to complete diagnostic procedures including a cardiac biopsy. Supportive care (e.g., oxygen). If no improvement within 3 to 5 days despite IV methylprednisolone at 2 to 4 mg/kg/day, promptly start immunosuppressive therapy such as TNF inhibitors (e.g., infliximab at 5 mg/kg every 2 weeks). Caution: It is important to rule out sepsis and refer to infliximab label for general guidance before using infliximab. Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, or anti-PJP treatment (refer to current NCCN guidelines for treatment of cancer- related infections [Category 2B |
| indicated (e.g.,<br>continuous IV<br>therapy or | discontinue study<br>drug/study regimen. | recommendation]). <sup>a</sup> |

mechanical hemodynamic support))

Myositis/Polymyositis
("Poly/myositis")

Date 10/08/2018

**Any Grade** 

#### General Guidance

#### For Any Grade:

- Monitor patients for signs and symptoms of poly/myositis. Typically, muscle weakness/pain occurs in proximal muscles including upper arms, thighs, shoulders, hips, neck and back, but rarely affects the extremities including hands and fingers; also difficulty breathing and/or trouble swallowing can occur and progress rapidly. Increased general feelings of tiredness and fatigue may occur, and there can be new-onset falling, difficulty getting up from a fall, and trouble climbing stairs, standing up from a seated position, and/or reaching up.
- If poly/myositis is suspected, a
   Neurology consultation should be
   obtained early, with prompt guidance
   on diagnostic procedures.
   Myocarditis may co-occur with
   poly/myositis; refer to guidance
   under Myocarditis. Given breathing
   complications, refer to guidance
   under Pneumonitis/ILD.
   Given possibility of an existent (but
   previously unknown) autoimmune
   disorder, consider Rheumatology
   consultation.
- Consider, as necessary, discussing with the study physician.
- Initial work-up should include clinical evaluation, creatine kinase, aldolase, LDH, BUN/creatinine, erythrocyte sedimentation rate or Creactive protein level, urine myoglobin, and additional laboratory work-up as indicated, including a number of possible rheumatological/antibody tests (i.e., consider whether a rheumatologist consultation is indicated and could guide need for rheumatoid factor, antinuclear antibody, anti-smooth muscle, antisynthetase [such as anti-Jo-1], and/or signal-recognition particle antibodies). Confirmatory testing may include electromyography, nerve conduction

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

studies, MRI of the muscles, and/or a muscle biopsy. Consider Barium swallow for evaluation of dysphagia or dysphonia.

Patients should be thoroughly evaluated to rule out any alternative etiology (e.g., disease progression, other medications, or infections).

#### Grade 1

(mild pain)

- No dose modifications.

#### For Grade 1:

- Monitor and closely follow up in 2 to 4 days for clinical symptoms and initiate evaluation as clinically indicated.
- Consider Neurology consult.
- Consider, as necessary, discussing with the study physician.

## For Grade 2:

- Monitor symptoms daily and consider hospitalization.
- Obtain Neurology consult, and initiate evaluation.
- Consider, as necessary, discussing with the study physician.
- If clinical course is rapidly progressive (particularly if difficulty breathing and/or trouble swallowing), promptly start IV methylprednisolone 2 to 4 mg/kg/day systemic steroids along with receiving input from Neurology consultant
- If clinical course is not rapidly progressive, start systemic steroids (e.g., prednisone 1 to 2 mg/kg/day PO or IV equivalent); if no improvement within 3 to 5 days, continue additional work up and start treatment with IV methylprednisolone 2 to 4 mg/kg/day
- If after start of IV methylprednisolone at 2 to 4 mg/kg/day there is no improvement within 3 to 5 days, consider start of immunosuppressive therapy such as TNF inhibitors (e.g., infliximab at 5 mg/kg every 2 weeks). Caution: It is important to rule out sepsis and refer to infliximab label for general guidance before using infliximab.
- Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, or anti-PJP

# Grade 2

(moderate pain associated with weakness; pain limiting instrumental activities of daily living [ADLs]) Hold study drug/study regimen dose until resolution to Grade ≤1.

Permanently
 discontinue study
 drug/study regimen if
 it does not resolve to
 Grade ≤1 within 30
 days or if there are
 signs of respiratory
 insufficiency.

Date 10/08/2018

#### Grade 3 or 4

(pain associated with severe weakness; limiting self-care ADLs)

# For Grade 3: Hold study drug/study

regimen dose until
resolution to Grade ≤1.

Permanently discontinue
study drug/study regimen
if Grade 3 imAE does not
resolve to Grade ≤1
within 30 days or if there
are signs of respiratory
insufficiency.

#### For Grade 4:

 Permanently discontinue study drug/study regimen. treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]).<sup>a</sup>

# For Grade 3 or 4 (severe or life-threatening events):

- Monitor symptoms closely; recommend hospitalization.
- Obtain Neurology consult, and complete full evaluation.
- Consider, as necessary, discussing with the study physician.
- Promptly start IV
  methylprednisolone 2 to 4 mg/kg/day
  systemic steroids <u>along with</u>
  receiving input from Neurology
  consultant.
- If after start of IV methylprednisolone at 2 to 4 mg/kg/day there is no improvement within 3 to 5 days, consider start of immunosuppressive therapy such as TNF inhibitors (e.g., infliximab at 5 mg/kg every 2 weeks). Caution: It is important to rule out sepsis and refer to infliximab label for general guidance before using infliximab.
- Consider whether patient may require IV IG, plasmapheresis.
- Once the patient is improving, gradually taper steroids over ≥28 days and consider prophylactic antibiotics, antifungals, or anti-PJP treatment (refer to current NCCN guidelines for treatment of cancerrelated infections [Category 2B recommendation]).<sup>a</sup>

<sup>a</sup>ASCO Educational Book 2015 "Managing Immune Checkpoint Blocking Antibody Side Effects" by Michael Postow MD.
 <sup>b</sup>FDA Liver Guidance Document 2009 Guidance for Industry: Drug Induced Liver Injury – Premarketing Clinical Evaluation.
 AChE Acetylcholine esterase; ADL Activities of daily living; AE Adverse event; ALP Alkaline phosphatase test; ALT
 Alanine aminotransferase; AST Aspartate aminotransferase; BUN Blood urea nitrogen; CT Computed tomography;
 CTCAE Common Terminology Criteria for Adverse Events; ILD Interstitial lung disease; imAE immune-mediated adverse event; IG Immunoglobulin; IV Intravenous; GI Gastrointestinal; LFT Liver function tests; LLN Lower limit of normal; MRI Magnetic resonance imaging; NCI National Cancer Institute; NCCN National Comprehensive Cancer Network; PJP *Pneumocystis jirovecii* pneumonia (formerly known as *Pneumocystis carinii* pneumonia); PO By mouth;
 T3 Triiodothyronine; T4 Thyroxine; TB Total bilirubin; TNF Tumor necrosis factor; TSH Thyroid-stimulating hormone; ULN Upper limit of normal.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

# **Infusion-Related Reactions**

| Severity Grade of<br>the Event (NCI<br>CTCAE<br>version 4.03) | Dose Modifications | Toxicity Management |
|---|---|---|
| Any Grade | General Guidance | For Any Grade: - Manage per institutional standard at the discretion of investigator. - Monitor patients for signs and symptoms of infusion-related reactions (e.g., fever and/or shaking chills, flushing and/or itching, alterations in heart rate and blood pressure, dyspnea or chest discomfort, or skin rashes) |
| | | and anaphylaxis (e.g., generalized urticaria, angioedema, wheezing, hypotension, or tachycardia). |
| Grade 1 or 2 | For Grade 1: | For Grade 1 or 2: |
| | The infusion rate of study drug/study regimen may be decreased by 50% or temporarily interrupted until resolution of the event. | <ul> <li>Acetaminophen and/or antihistamines may be administered per institutional standard at the discretion of the investigator.</li> <li>Consider premedication per institutional standard prior to subsequent doses.</li> <li>Steroids should not be used for routine premedication of Grade ≤2 infusion reaction</li> </ul> |
| | For Grade 2: | • |
| | The infusion rate of study drug/study regimen may be decreased 50% or temporarily interrupted until resolution of the event. | |
| | Subsequent infusions may be given at 50% of the initial infusion rate. | |
| Grade 3 or 4 | For Grade 3 or 4: | For Grade 3 or 4: |
| | Permanently discontinue study drug/study regimen. | <ul> <li>Manage severe infusion-related reactions per<br/>institutional standards (e.g., IM epinephrine,<br/>followed by IV diphenhydramine and<br/>ranitidine, and IV glucocorticoid).</li> </ul> |

CTCAE Common Terminology Criteria for Adverse Events; IM intramuscular; IV intravenous; NCI National Cancer Institute.

Clinical Study Protocol Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

## **Non-Immune-Mediated Reactions**

| Severity Grade of the<br>Event (NCI CTCAE<br>version 4.03) | Dose Modifications | Toxicity Management |
|---|---|---|
| Any Grade | Note: Dose modifications are not required for AEs not deemed to be related to study treatment (i.e., events due to underlying disease) or for laboratory abnormalities not deemed to be clinically significant. | Treat accordingly, as per institutional standard. |
| Grade 1 | No dose modifications. | Treat accordingly, as per institutional standard. |
| Grade 2 | Hold study drug/study regimen until resolution to ≤Grade 1 or baseline. | Treat accordingly, as per institutional standard. |
| Grade 3 | Hold study drug/study regimen until resolution to ≤Grade 1 or baseline. | Treat accordingly, as per institutional standard. |
| | For AEs that downgrade to \(\leq\)Grade 2 within 7 days or resolve to \(\leq\)Grade 1 or baseline within 14 days, resume study drug/study regimen administration. Otherwise, discontinue study drug/study regimen. | |
| Grade 4 | Discontinue study drug/study regimen (Note: For Grade 4 labs, decision to discontinue should be based on accompanying clinical signs/symptoms, the Investigator's clinical judgment, and consultation with the Sponsor.). | Treat accordingly, as per institutional standard. |

Note: As applicable, for early phase studies, the following sentence may be added: "Any event greater than or equal to Grade 2, please discuss with Study Physician."

AE Adverse event; CTCAE Common Terminology Criteria for Adverse Events; NCI National Cancer Institute.

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4

Date 10/08/2018

## APPENDIX B: DURVALUMAB DOSE CALCULATIONS

## **Durvalumab Dosing**

The durvalumab dosing should be done depending on subject weight (if subject is < 30kg) at 20 mg/kg:

- 1. Cohort dose: X mg/kg
- 2. Subject weight: Y kg
- 3. Dose for subject: XY mg =  $X (mg/kg) \times Y (kg)$
- 4. Dose to be added into infusion bag:

Dose 
$$(mL) = XY mg / 50 (mg/mL)$$

where 50 mg/mL is durvalumab nominal concentration

The corresponding volume of durvalumab should be rounded to the nearest tenth mL (0.1 mL). Dose adjustments for each cycle only needed for greater than 10% change in weight.

5. The theoretical number of vials required for dose preparation is the next greatest whole number of vials from the following formula:

Number of vials = Dose (mL) / 10 (mL/vial)

# **Example:**

- 1. Cohort dose: 10 mg/kg
- 2. Subject weight: 30 kg
- 3. Dose for subject:  $300 \text{ mg} = 10 \text{ (mg/kg)} \times 30 \text{ (kg)}$
- 4. Dose to be added into infusion bag:

Dose 
$$(mL) = 300 \text{ mg} / 50 \text{ (mg/mL)} = 6.0 \text{ mL}$$

5. The theoretical number of vials required for dose preparation:

Number of vials = 
$$6.0 \text{ (mL)} / 10.0 \text{ (mL/vial)} = 1 \text{ vials}$$

Drug Substance Durvalumab (Medi4736)

Study Number MCC 18788/MCC18788/ESR-15-11326

Edition Number 1.9.4
Date 10/08/2018

# **APPENDIX C**

Schedule of study procedures: follow-up for subjects who have discontinued durvalumab due to toxicity in the absence of confirmed progression of disease

| | Time Since Last Dose of durvalumab | | | | | | |
|---|---|---|---|---|---|---|---|
| Evaluation | Day (±3) | | Months (±1 week) | | | | |
| | 30 | 2 | 3 | 5 | 7 | 9 | 12 |
| Physical examination <sup>a</sup> | Х | | | | | | |
| Vital signs (temperature, respiratory rate, blood pressure, pulse) | х | | | | | | |
| Weight | X | | | | | | |
| AE/SAE assessment | X | X | X | | | | |
| Concomitant medications | X | X | X | | | | |
| < <world health="" organisation="">&gt; &lt;<ecog>&gt; performance status<sup>b</sup></ecog></world> | Х | X | X | | | | |
| Subsequent anti-cancer therapy | X | X | X | X | X | X | X |
| Survival status: phone contact with subjects who refuse to return for evaluations and agree to be contacted | | X | X | X | X | X | X |
| Urine hCG or serum βhCG | X | | | | | | |
| Hematology | Х | X | X | | | | |
| Serum chemistry | X | X | X | | | | |
| Thyroid function tests (TSH, and fT3 and fT4) <sup>c</sup> | х | | | | | | |
| Tumour assessment (CT or MRI) | At the discretion of treating physician, which is not indicated until the localized bladder cancer progressed to the muscle invasive stage (T2 or above) X | | | | | | |

a Full physical exam

PS to be collected if available at the 2 monthly calls to obtain subsequent anti-cancer therapy and survival status

Free T3 and free T4 will only be measured if TSH is abnormal. They should also be measured if there is clinical suspicion of an adverse event related to the endocrine system.

Date 10/08/2018

# **APPENDIX D**

Schedule of study procedures: follow-up for subjects who have discontinued durvalumab treatment due to confirmed progression of disease at the investigator discretion

| | Time Since Last Dose of durvalumab | | | | | | |
|---|---|---|---|---|---|---|---|
| Evaluation | Day (±3) | | Months (±1 week) | | | | |
| | 30 | 2 | 3 | 5 | 7 | 9 | 12 |
| Physical examination <sup>a</sup> | X | | | | | | |
| Vital signs (temperature, respiratory rate, blood pressure, pulse) | X | | | | | | |
| Weight | X | | | | | | |
| AE/SAE assessment | X | X | X | | | | |
| Concomitant medications | X | X | X | | | | |
| < <world health="" organisation="">&gt;<br/>&lt;<ecog>&gt; performance status<sup>b</sup></ecog></world> | X | X | X | | | | |
| Subsequent anti-cancer therapy | X | X | X | X | X | X | X |
| Survival status: phone contact with subjects who refuse to return for evaluations and agree to be contacted | | X | X | X | X | X | X |
| Urine hCG or serum βhCG | X | | | | | | |
| Hematology | X | X | X | | | | |
| Serum chemistry | X | X | X | | | | |
| Thyroid function tests (TSH, and fT3 and fT4) <sup>c</sup> | X | | | | | | |
| Tumour assessment (CT or MRI) | At the discretion of treating physician, which is not indicated until the localized bladder cancer progressed to the muscle invasive stage (T2 or above) X | | | | | | |

a Full physical exam

PS to be collected if available at the 2 monthly calls to obtain subsequent anti-cancer therapy and survival status

Free T3 and free T4 will only be measured if TSH is abnormal. They should also be measured if there is clinical suspicion of an adverse event related to the endocrine system.